

# Protocol for non-interventional studies based on existing data

| Document number: c03856813-11 | |
|---|---|
| BI Study number: 1245.97 | |
| BI Investigational Product(s): Jardiance® (empagliflozin), Synjardy® (empagliflozin/metformin hydrochloride) | |
| Title: | Post-authorisation safety study to assess the risk of urinary tract malignancies in relation to empagliflozin exposure in patients with type 2 diabetes: a multi-database European study |
| Protocol version identifier: | 8.0 |
| Date of last version of protocol: 07 July 2022 | |
| PASS: | Yes |
| EU PAS register number: | EUPAS16424 |
| Active substance: | A10BK03 empagliflozin, A10BD20 metformin and empagliflozin |
| Medicinal product: | Jardiance, Synjardy |
| <b>Product reference:</b> | EMEA/H/C/002677, EMEA/H/C/003770 |
| Procedure number: | EMEA/H/C/002677/MEA; EMEA/H/C/003770/MEA |
| Joint PASS: | No |
| Research question and objectives: The aim of the study is to assess the risk of urinary trace malignancies in patients initiating empagliflozin compatients initiating a DPP-4 inhibitor. | |

| Countries of study: | The United Kingdom, Sweden, and Finland |
|---|---|
| Authors: | |
| Marketing authorisation holder(s): | |
| MAH contact person: | |
| EU-QPPV: | |
| Signature of EU-<br>QPPV: | The signature of the EU-QPPV is provided electronically |
| Date: | 17 May 2023 |

## **Proprietary confidential information**

© 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

## **TABLE OF CONTENTS**

| T | ITLE PAGE | | 1 |
|---|---|---|---|
| Τ. | ABLE OF CO | NTENTS | 3 |
| L | IST OF TABI | LES | 6 |
| L | IST OF FIGU | RES | 7 |
| 1. | LIST OF A | ABBREVIATIONS | 8 |
| 2. | RESPONS | SIBLE PARTIES | 10 |
| 3. | ABSTRAC | CT | 11 |
| 4. | AMENDM | MENTS AND UPDATES | 21 |
| 5. | | NES | |
| 6. | RATIONA | ALE AND BACKGROUND | 28 |
| | 6.1<br>DIABETES 1 | EPIDEMIOLOGY OF URINARY TRACT MALIGNANCIES IN PATIENTS | 29 |
| | 6.1.1 and Swede | Incidence of urinary tract malignancies in the study population in the UK en observed in the fifth interim report of this study | |
| | 6.2<br>PATTERNS | EPIDEMIOLOGY OF DIABETES AND DIABETES TREATMENT IN THE UK | 31 |
| | 6.3<br>PATTERNS | EPIDEMIOLOGY OF DIABETES AND DIABETES TREATMENT IN SWEDEN AND FINLAND | 32 |
| | 6.4<br>INHIBITORS | RISK OF BLADDER CANCER IN PREVIOUS TRIALS OF SGLT-2 | 32 |
| | 6.5 | RATIONALE FOR THE PROTOCOL AMENDMENT | 32 |
| 7. | RESEARC | CH QUESTION AND OBJECTIVES | 34 |
| 8. | RESEARC | CH METHODS | .35 |
| | 8.1 | STUDY DESIGN | .35 |
| | 8.2 | SETTING | .36 |
| | 8.2.1 | Study populations | .36 |
| | 8.2.2 | Study period | 37 |
| | 8.2.3 | Index date | 37 |
| | 8.2.4 | Baseline and look-back (pre-index) period | 37 |
| | 8.2.5 | Inclusion and exclusion criteria. | 37 |
| | 8.3 | VARIABLES | 38 |
| | 8.3.1 | Exposures | 39 |
| | 8.3.2 | Outcomes | .41 |

| | 8.3.2.1 | Primary outcomes | 41 |
|---|---|---|---|
| | 8.3.3 | Covariates | 42 |
| | 8.3.4 | Censoring of follow-up time | |
| | 8.3.5 | | |
| 0 | | Follow-up time | |
| 8. | | DATA SOURCES | |
| | 8.4.1 | The United Kingdom Clinical Practice Research Datalink (CPRD) | |
| | 8.4.2 | Swedish national registries | |
| | 8.4.3 | Finnish data sources | |
| _ | 8.4.4 | Additional potential data sources | |
| 8. | | STUDY SIZE | |
| 8. | | DATA MANAGEMENT | |
| 8. | .7 | DATA ANALYSIS | |
| | 8.7.1 | Main analysis | |
| | 8.7.1.1 | Matching at index date | 63 |
| | 8.7.1.2 | As-treated (AT) analysis | 64 |
| | 8.7.1.3 | Population summary and descriptive analyses | 65 |
| | 8.7.1.4 | Comparative analyses | 65 |
| | 8.7.1.5 | Variable selection | 66 |
| | 8.7.1.6 | Monitoring of accrual of empagliflozin users | 66 |
| | 8.7.1.7 | Handling of missing data | 67 |
| 8. | .8 | QUALITY CONTROL | 69 |
| 8. | .9 | LIMITATIONS OF THE RESEARCH METHODS | 70 |
| | 8.9.1 | Bias | 71 |
| | 8.9.2 | Generalizability | 71 |
| 9. | PROTECT | ΓΙΟΝ OF HUMAN SUBJECTS | 73 |
| 10. | MANA | GEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE | |
| REA | ACTIONS | | 74 |

| 11. | PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESU | ULTS .75 |
|------|---------------------------------------------------------|----------|
| 12. | REFERENCES | 76 |
| 12.1 | PUBLISHED REFERENCES | 76 |
| 12.2 | UNPUBLISHsED REFERENCES | 80 |
| 13. | ANNEXURE | 81 |
| AN. | NEX 1. LIST OF STAND-ALONE DOCUMENTS | 81 |
| AN. | NEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS | 82 |
| AN. | NEX 3. READ CODES TO IDENTIFY TYPE 2 DIABETES | 88 |
| AN | NEX 4. CODES TO IDENTIFY EXPOSURE VARIABLES | 104 |
| AN | NEX 5. CODES TO IDENTIFY THE OUTCOME VARIABLES | 107 |
| AN | NEX 6. COVARIATES TO BE CONSIDERED FOR INCLUSION IN THE | |
| PRO | OPENSITY SCORE MODEL. | 109 |
| SIGN | ATURE | 111 |

## LIST OF TABLES

| Table 1. | Crude incidence rates per 100,000 person-years for urinary tract cancers, Nordic countries 2013 and the UK 2012 | 29 |
|---|---|---|
| Table 2. | Patient counts by Glucose Lowering Medication category in the UK, | |
| Table 2 | Sweden, and Finland | |
| Table 3. | Exposure definitions for primary and secondary analyses | <u>40</u> |
| Table 4. | Baseline covariates to be considered for inclusion alternatively or simultaneously in primary, secondary, and further analyses | 12 |
| Table 5. | Minimum data requirements and data availability for the UK and the national registries in Sweden and Finland | |
| Table 6. | Observed and expected number of patients eligible for inclusion in the study population, by study drug group (including fixed-dose combinations with metformin), by study country and overall, using an arithmetic growth | . <u>55</u> |
| Table 7. | Power for different effect sizes for single-country analyses based on Cox models with a type 1 error probability of 5%, given country-level observed incidence rates, expected numbers of empagliflozin initiators, expected follow-ups, and expected matching ratios. | . 57 |
| Table 8. | Power of meta-analyses for a type 1 error probability of 5% for different effect sizes, given country-level observed incidence rates, expected number of empagliflozin initiators, expected average follow-ups, and expected matching ratios. | |
| Table 9. | Minimum detectable effect sizes (Hazard Ratios) given country-level observed incidence rate, expected sample sizes, expected average follow-ups, and matching ratios for single-country analyses and meta-analyses for a type 1 error probability of 5%. | |
| Table 10. | Required sample sizes in each study country to estimate different effect sizes for the three primary endpoints in the single-country analyses with at least 80% power and a type 1 error probability of 5%, given country-level incidence rates, expected average follow-ups, and expected matching ratios. | |
| Table 11. | Required sample sizes in each study country to estimate different effect sizes for the three primary endpoints in the meta- analyses with at least 80% power and a type 1 error probability of 5%, given country-level incidence rates, expected average follow-ups, and expected matching ratios | |
| Table 12. | Required follow-up time (years) to achieve 80% power in country-level analyses with a type 1 error probability of 5% for different effect sizes for the three primary endpoints given country-level observed incidence rates, expected sample sizes, and expected matching ratios | |
| Table 13. | Required follow-up time (years) in each study country to achieve 80% power for the meta-analysis with a type 1 error probability of 5% for different effect sizes for the three primary endpoints given country-level observed incidence rates, expected sample sizes, and expected matching ratio | |

## Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1245.97


c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF FIGURES

| Figure 1 | Discontinuation of index drug due to stopping of index drug or switching of |
|---|---|
| | index drug. In the primary analysis follow-up is censored at treatment |
| | discontinuation |

## 1. LIST OF ABBREVIATIONS

AT As-treated analysis

ATC Anatomical Therapeutic Chemical Classification System

AvoHILMO Register of primary health care visits

BI Boehringer Ingelheim International GmbH

BMI Body mass index

CI Confidence interval

COPD Chronic obstructive pulmonary disease

CPRD Clinical Practice Research Datalink

CV Cardiovascular

DDD Defined daily dose

DPP-4 Dipeptidyl peptidase-4

eGFR Estimated glomerular filtration rate

EMA European Medicines Agency

EMR Electronic medical record

ENCePP European Network of Centres for Pharmacoepidemiology and

Pharmacovigilance

EU European Union

FDA Food and Drug Administration

GLP-1 Glucagon-like peptide-1

GP General practitioner

GPP Good Pharmacoepidemiology Practices

GPV Good Pharmacovigilance Practices

HbA1c Glycated haemoglobin A1c HES Hospital Episode Statistics

HF Heart failure

HILMO Care register for health care

HR Hazard ratio

HUS Helsinki University Hospital region ICD-10 International classification of diseases

IPTW Inverse-probability of treatment weights

## **Boehringer Ingelheim**

# Protocol for non-interventional studies based on existing data

BI Study Number 1245.97 c03856813-11


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

ITT Intention-to-treat analysis

MI Myocardial infarction

MSM Marginal structural model

NCC Nested case-control

NHS National Health Service

NSAID Non-steroidal anti-inflammatory drugs

ONS Office for National Statistics

PASS Post-safety study

PH Proportional hazards

PID Personal identification number

PS Propensity score

PSUR Periodic Safety Update Report

PY Person-years

RMP Risk management plan

RR Relative risk

SEAP Statistical/Epidemiological Analysis Plan

SGLT-2 Sodium glucose co-transporter-2

SID Study identification number

SIR Standardized incidence ratio

T2D Type 2 diabetes mellitus

THIN The Health Improvement Network database

UK United Kingdom

US United States
UT Urinary tract

UTI Urinary tract infection

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2. RESPONSIBLE PARTIES





## **Sponsor**

Boehringer Ingelheim International GmbH

The study investigators at Company) share responsibility with Boehringer Ingelheim International GmbH (BI) for the design of the study. The investigators are responsible for conducting the study in a manner that meets regulatory standards, conducting analyses, and preparing scientific reports. The study shall be conducted as described in the approved protocol. The authors will not develop or implement any deviation or change to the protocol without prior review by BI.

The financial sponsor of this study is BI. The sponsor is responsible to assure study progress. BI is also responsible for communicating with the European Medicines Agency (EMA) (called 'the agency') about the study protocol, the progress of the study, and study results.

# 3. ABSTRACT

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of the finished medicinal product: Jardiance®, Synjardy | | | |
| Name of active ingr<br>Empagliflozin (A10I<br>Metformin and empa | | | |
| Protocol date: | Study number/ Document number: | Version/Revision: | Version/Revision date: |
| 16-Sep-2015 | 1245.97 / c03856813-10 | 8.0 | 17-May-2023 |
| Title of study: | | study to assess the risk of urinexposure in patients with type 2 | |
| Rationale and background: Empagliflozin is an oral ble co-transporter-2 (SGLT-2) excretion of glucose and he 2 diabetes. As a part of the risk manage hydrochloride agreed upon authorisation safety study malignancies in patients dipeptidyl peptidase-4 (DF this study, a feasibility as Research Datalink (CPRI Statistics (HES), and Offic United Kingdom (UK) as performed with the aim to assess, for each potential information for urinary the registries, mortality registricountries, the UK (CPRD 2019. In order to increase initiating the study drugs a risk of malignancies, the stand Finnish national registro.), CPRD Aurum was income | | ood glucose lowering drug belon ) inhibitor class. SGLT-2 inhi- elp lower elevated blood glucose gement plans for empagliflozin and on by the European Medicines (PASS) will be performed to assinitiating empagliflozin, compagned inhibitors. Prior to the deverous essessment of three databases in the potential for the compagned inhibitors. Prior to the deverous effect of National Statistics (ONS) and data with potential for the for National Statistics (ONS) and the national registers in Solution detail the minimum data required data source, the data quality, ract malignancies, and possibilities, and other data sources. Initiate GOLD) and Sweden, with following the accumulated patient year as well as accounting for the longudy follow-up was first extended ters were included. In this version further increasing the sample size increasing study power. | ibitors promote the renal levels in patients with type and empagliflozin/metformin Agency (EMA), a postess the risk of urinary tract ared to patients initiating lopment of the protocol for Europe (Clinical Practice linkage (Hospital Episode mortality statistics) in the sweden and Finland) was ements for the study and to completeness of recorded ty of linkage with cancer lly, this study included two w-up until 31st December, sand number of patients ag latency period related to until 31st December, 2020 on of the protocol (Version ded to 31st December, 2021 |

# Protocol for non-interventional studies based on existing data BI Study Number 1245.97

c03856813-11

| Name of compan | ıy: | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of the finished medicinal product: Jardiance®, Synjardy | | | |
| Name of active ingre<br>Empagliflozin (A10E | BK03) | | |
| Metformin and empa | · | | |
| 16-Sep-2015 | 1245.97 / c03856813-10 | 8.0 | 17-May-2023 |
| Research question and objectives: | | o assess the risk of urinary trac<br>ee or fixed-dose combination) con | |
| | urinary tract cance patients initiating inhibitor (ii) To estimate the af empagliflozin con (iii) To estimate the af | estimate the adjusted hazard ratios (aHRs) and incidence rates (IRs) of all hary tract cancers (bladder, renal and other urinary tract cancers) in tents initiating empagliflozin compared to patients initiating a DPP-4 libitor estimate the aHRs and IRs of bladder cancer in patients initiating pagliflozin compared to patients initiating a DPP-4 inhibitor estimate the aHRs and IRs of renal cancer in patients initiating pagliflozin compared to patients initiating a DPP-4 inhibitor | |
| | To estimate the a cancers, bladder c a. increasin b. dosage o empaglif | e the aHRs and IRs of each primary outcome (all urinary dder cancer, renal cancer) with respect to: creasing cumulative dosage of empagliflozin exposure sage of empagliflozin prescribed per use (e.g., 10mg vs 25 apagliflozin) he since first dose of empagliflozin exposure | |

| Name of same | | | |
|---|---|---|---|
| Name of company: | | | |
| Boehringer Ingel | heim | | |
| Name of the finished medicinal product: Jardiance®, Synjardy | | | |
| Name of active ingr<br>Empagliflozin (A10) | | | |
| Metformin and empa | ngliflozin (A10BD20) | | |
| 16-Sep-2015 | 1245.97 / c03856813-10 | 8.0 | 17-May-2023 |
| Study design: | This is a non-interventional, comparative, cohort safety study based on European healthcare databases. The databases for this study are constructed from linked prescription, hospital, general practitioner, cancer and death registration records. The study will use an "incident users" design and compare new users of empagliflozin to new users of DPP-4 inhibitors. The index date will be defined as the date on which each identified new user receives the index prescription for empagliflozin, or a DPP-4 inhibitor. Follow-up will start 6 months after the index date (12 months in sensitivity analyses) to account for an empirical induction/promotion period. To minimize channelling bias, individuals will be matched with similar treatment and clinical history at index date by deriving propensity scores (PS). PS-matched cohorts will be derived for the comparison from the study base by matching patients who initiate empagliflozin with patients who initiate DPP-4 inhibitors at index date. To further gain power, the highest possible matching ratio in each country-level dataset will be used. This will be implemented using a variable ratio approach in all countries, where exposed patients are matched to as many control patients as possible, up to a maximum of 3 matched controls. Thus, an observational cohort is constructed to study the risk of urinary tract cancer among the two treatment groups. Depending on sample size, combination exposures with metformin will be accounted for through separate PS, stratification, or | | |

| Name of compar | ny: | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of the finished medicinal product: Jardiance®, Synjardy | | | |
| Name of active ingr<br>Empagliflozin (A10E<br>Metformin and empa | | | |
| 16-Sep-2015 | 1245.97 / c03856813-10 | 8.0 | 17-May-2023 |
| Population: | Aurum in the UK and patic have purchased at least of during the study period 20 or DPP-4 inhibitor fixed-d. Index date: Date of first p during follow-up (2014-2 inhibitor fixed-dose combit The study population will following inclusion and ex Inclusion criteria: Diagnosis of type Age over 18 years At least 1 year of least 1 year of condindex date Exclusion criteria: Patients with any date Diagnosis of type Use of any SGLT dose combination Use of fixed-dose Diagnosis of end stage ren | oad study population will include all patients from CPRD GOLD and CPRD in the UK and patients in the nationwide registers in Sweden and Finland, who urchased at least one prescription of empagliflozin, or DPP-4 inhibitor drugs the study period 2014-2020 (2021 for CPRD). Patients initiating empagliflozin, or 4 inhibitor fixed-dose combinations with metformin will be included. **date: Date of first purchase/prescription of empagliflozin, or a DPP-4 inhibitor follow-up (2014-2020; 2014-2021 for CPRD). Patients initiating DPP-4 or fixed-dose combinations with metformin will also be included. **udy population will be selected from the broad study population with the ing inclusion and exclusion criteria: **Diagnosis of type 2 diabetes (T2D) **Age over 18 years at index date At least 1 year of membership in the database prior to index date; in CPRD, at least 1 year of continuous up-to-standard registration in the CPRD prior to the index date ion criteria: **Patients with any cancer (excluding non-melanoma skin cancer) prior to index | |
| Variables: | Outcome variables: | | |

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of the finished medicinal product: Jardiance®, Synjardy | | | |
| Name of active ingre<br>Empagliflozin (A10E | | | |
| Metformin and empa | gliflozin (A10BD20) | | |
| 16-Sep-2015 | 1245.97 / c03856813-10 | 8.0 | 17-May-2023 |
| | | | agliptin, vildagliptin, or ed-dose combinations with drugs prior to index date is 10mg vs 25 mg), and for as variables for exact or in the risk set definition in rive inverse-probability of is (MSMs) and/or model todes recorded prior to the fied below. ex date, length of available ducose lowering medication etes medications) HbA1c value) |
| | <ul> <li>BMI, smoking, alcohol use (closest to index date)</li> <li>Additional covariates will be included according to data availability are, such as socioeconomic position and laboratory measurements.</li> </ul> | | |

## Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1245.97


c03856813-11

| N. 0 | | | |
|---|---|---|---|
| Name of company: | | | |
| Boehringer Ingell | heim | | |
| Name of the finished medicinal product: Jardiance®, Synjardy | | | |
| Name of active ingr<br>Empagliflozin (A10E<br>Metformin and empa | | | |
| Protocol date: | Study number/ | Version/Revision: | Version/Revision date: |
| 16-Sep-2015 | <b>Document number:</b> 1245.97 / c03856813-10 | 8.0 | 17-May-2023 |
| Data sources: | database for each country of The UK: CPRD GOLD (Outpatient data, and Adm Sweden: The following not National Patient Register, Register, the Causes of Longitudinal integration data Finland: The following not Finnish prescription regists for health care (HILMO), the Finnish cancer regists (EMR) databases will be a Initially, the country-level level estimates will be produce as narrow confider If patient numbers accument. | re country-specific data sources familia be constructed. and CPRD Aurum optionally itted Patient Care data), and ONS ationwide population-based regist the Swedish Prescribed Drug Re Death Register, the National Database for health insurance and I ationwide population-based register/the registry for reimbursed methe Register of primary health carer. Additionally, four regional coessed to obtain information on datasets will be analysed separt ooled using meta-analysis technice intervals (CI) as possible. | complemented with HES is mortality sources. Sters will be accessed: The gister, the Swedish Cancer biabetes Register, and the abor market studies. Sters will be accessed: the dications, the Care register the visits (AvoHILMO), and electronic medical record laboratory measures. ately. Thereafter, country-niques to gain power and |

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingell | neim | | |
| Name of the finish product: Jardiance®, Synja | | | |
| Name of active ingr<br>Empagliflozin (A10E | BK03) | | |
| Metformin and empa | gliflozin (A10BD20) | | |
| 16-Sep-2015 | 1245.97 / c03856813-10 | 8.0 | 17-May-2023 |
| Study size: | the treatment of T2D to in Finland. Study-size and pot the primary outcomes. On approximately 18,000 emp Swedish databases. Howe monitoring report (2019), approximately 25,000 emp Further, additional 38,000 of Finnish databases, for a Updated estimates in the empagliflozin initiators we GOLD, Sweden, and Finlatof CPRD-Aurum and the CPRD databases suggest the for inclusion across all three initiating DPP-4 inhibitors would be 1:3 in UK-CPRD Power to detect relative ristor each of the study outco to empagliflozin eligible for 16,887 in UK-CPRD (GOI and the observed IRs of ur country-level study popula 111.5, 66.7, 26.5 per 100 of Finland: 161.5, 86.8, 71.6 bladder cancer and renal car comparison between empa power at the meta-analysis | ren by the uptake of empagliflozing prove glycaemic control in adult ower computations were carried of Driginally, it was expected the agliflozin-treated patients will active, based on the conservative the expected sample size was his pagliflozin initiators eligible for patients were expected by the encetotal of approximately 78,000 by fifth interim report (2021) indicate expected to be eligible for including by the end 2020. New estimative extension of the study period to that a total of 67,490 empagliflozing extension of the study period to the expected to be eligible for including the extension of the study period to the extension of the study for each the expected number inclusion in the study for each the expected number inclusion in the study for each the expected in the fifth interpolation as reported in the fifth interpolation as reported in the fifth interpolation. Power calculations perfor gliflozin users and DPP-4 inhibitately for detecting a hazard ratio of the expected provides and the expective power would be 97.0%. | Its in the UK, Sweden, and but for the meta-analysis of that by the end of 2019, but mulate in the CPRD and the estimates from the third igher than anticipated with for inclusion in the study. If of 2020 with the inclusion the end of the study period. It attends that a total of 57,000 assion in the study in CPRD-attends including the inclusion of the end of 2021 for both in initiators could be eligible served numbers of patients achievable matching ratios and. It the meta-analysis level, ber of individuals exposed country (approximately en, and 18,269 in Finland) or and renal cancer in the report (UK-CPRD: 3.0 per 100 000 PY; or urinary tract cancer, med for the primary tors indicated that the of 1.5 would be 93.6% |

## Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1245.97


c03856813-11

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingell | neim | | |
| Name of the finished medicinal product: Jardiance®, Synjardy | | | |
| Name of active ingr<br>Empagliflozin (A10E<br>Metformin and empa | | | |
| 16-Sep-2015 | 1245.97 / c03856813-10 | 8.0 | 17-May-2023 |
| | In addition, anticipated study sample size would ensure sufficient power for the meta-<br>analysis to detect the targeted effect size of $< 1.6$ for urinary tract cancers and bladder<br>cancer and the targeted effect size of $< 2.0$ for renal cancer, with 80% power under the<br>expected matching ratios in each study country. | | |
| | Results from the second and third interim analysis showed that not enough patients wi have accumulated in the UK CPRD or Swedish registers by the planned end of dat collection to reach the desired sample size. For this reason, the protocol was first amended to expand the study population by including data from the Finnish national registries and extend the study period until 31st December 2020. Following results from the fifth interim analysis, the protocol was further amended to also include the CPRI Aurum database and to extend the study period to the end of 2021 for both CPRI databases. | | |

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of the finished medicinal product: Jardiance®, Synjardy | | | |
| Name of active ingr<br>Empagliflozin (A10E<br>Metformin and empa | 3K03) | | |
| Protocol date: | Study number/<br>Document number: | Version/Revision: | Version/Revision date: |
| 16-Sep-2015 | 1245.97 / c03856813-10 | 8.0 | 17-May-2023 |
| Data analysis: | conducted in two stages: (exposure to empagliflozin aHR compared to those exposure to empagliflozin aHR compared to those exposure undefinitions of outcome, exposure undefinitions of outcome, exposure undefinition and presence of empagliflozin exposure undempagliflozin, and metfor compared with patients standard presented and adjusted) with the time-varying coverage of the page of the pa | will be presented for each exposurable Poisson regression approach (HRs) adjusted for relevant varial variate approach. The aHRs and I sestimates. Country-level estimates | d cohort by modelling the estimating the effect of al and other) cancers using respective IRs. Additional robustness of alternative is reduction of bias due to evaluate the current use of starting a combination of free combination) will be inhibitor and metformin. Etformin will be accounted the group and stratified by the Relative risks will be be be using the Cox's model Rs will be presented along |

## Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1245.97


c03856813-11

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingell | heim | | |
| Name of the finished medicinal product: Jardiance®, Synjardy | | | |
| Name of active ingr<br>Empagliflozin (A10I<br>Metformin and empa | | | |
| 16-Sep-2015 | 1245.97 / c03856813-10 | 8.0 | 17-May-2023 |
| Milestones: | Launch in the UK and Fi November 2014. Synjardy marketing authorisation in for review in September 2 version 4 in March 2019, a PAS register occurred in I protocol endorsement by the been monitored. Based on a decision will be made to interim report stage. Any d the length of the study per protocol amendment. Takin and Finnish data through I 2023. Analysis of CPRD 2023 and the final report | was granted EU marketing audinland was in August 2014; laurar (empagliflozin/metformin hydromay 2015. Protocol version 1 volume 2015, version 2 in February 2011 and protocol version 5.0 in Sep 2012 December 2016 (EUPAS16424) and EMA. The number of users in the available patient numbers and proceed with adjusted, treatment ecision based on the results of the riod or the use of other data souring into account the database lag December 2020 will be performed data through December 2021 will be finalised by Q2 2024. In data source were sent to EMA and the end of the total account the database lag December 2020 will be finalised by Q2 2024. | nch in Sweden took place ochloride) was granted EU was submitted to the EMA 6, version 3 in June 2016, 019. Registration in the EU and was updated following each treatment cohort have at the event rates observed, int-stratified analyses at the exinterim reports concerning rees will be approved via a gs, the analysis of Swedish d between Q3 2022 and Q3 ill be performed in Q3/Q4 Progress reports including |

## 4. AMENDMENTS AND UPDATES

| Amendment<br>number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 8.0 | 17 May<br>2023 | 5 | Update of planned date for final study report | Delayed CPRD<br>approval of study<br>collaborators agreement |
| 7.0 28 Jun<br>2022 | Multiple | Multiple | To include data from the Clinical Practice Research Datalink (CPRD) Aurum database in the study. | European Medicines Agency (EMA) requested to reconsider the inclusion of CPRD Aurum as an additional study database in the UK to capture as many CPRD UK patients as possible, increase the sample size, and improve the study power in this country. |
| | 28 June | Multiple | Study period extended until 31 <sup>st</sup> December 2021, for the CPRD (GOLD and Aurum). | To increase the sample size, and improve study power in the UK. |
| | 2022 | Multiple | To not include data from the Cancer registry from the United Kingdom (UK) in the study. | Data linkage for a sensitivity analysis (Section 8.7.2.3) is not available in time for the final report submission. |
| | | Multiple | To update the power calculations. | EMA requested to update the power calculations for the UK, taking into account the inclusion of CPRD Aurum as additional country-specific data source, and for Finland, taking into account that 1:2 matching ratio may be feasible in this country. |

| Amendment<br>number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| | | 8.7.1.4 | To briefly describe the appropriate statistical methods. | EMA requested to briefly describe the appropriate methods to combine results obtained from the main analysis performed in the different data sources, including the meta-analytical techniques such as the meta-analysis model and analysis and handling of heterogeneity or describe the process to identify the most appropriate method. |
| 6.0 | 26<br>January<br>2022 | Multiple | To not include data from the Clinical Practice Research Datalink (CPRD) Aurum database in the study. | The study will have adequate power to demonstrate a significant difference assuming the target hazard ratios with patients from the data sources mentioned in the study (i.e., national registers in Sweden and Finland and CPRD GOLD database). Therefore, additional data from the Aurum database is not needed. |

| Amendment<br>number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| | | | | Information on Aurum database was removed from this protocol. |
| | | Multiple | To use the highest possible matching ratio between initiators of empagliflozin and (dipeptidyl peptidase-4) DPP-4 inhibitors. | It was observed in the last interim report that there were not enough patients for 1:3 matching in Finland and Sweden. Therefore, 1:1 or highest possible matching ratio will be used in each country. |
| | | Multiple | To remove sodium glucose cotransporter-2 (SGLT-2) inhibitors as a comparison group from the study analyses. | It was observed in the last interim report that the yearly number of patients initiating SGLT-2 inhibitors other than empagliflozin decreased during the study period (2014-2020). The total number of SGLT-2 inhibitors was considerably lower than that of empagliflozin initiators (a 1:1 matching cannot be performed), therefore only patients initiating DPP-4 inhibitors will be used as a primary comparison group. |
| | | | | _ |

| Amendment<br>number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| | | 8.7 | Meta-Analysis | Data from Finland and Sweden cannot be transferred out of the country of origin. Therefore, pooling of all data and pooled analyses cannot be conducted. Information on pooled analyses was removed and instead meta-analysis was added to the protocol where relevant. |
| | | 8.4.3 | Findata | In Finland, all the data will be delivered to and analyzed in the remote access server environment provided by the national permit authority Findata. The data holders will extract the relevant data and deliver it to Findata for pseudonymization. |
| | | Multiple | Other minor updates. | To align updates holistically. |
| | Multiple | Inclusion of new study country, Finland. | To increase of the size of the patient population. | |
| 5.0 | 23<br>August<br>2019 | Multiple | Using DPP-4 inhibitors as the primary comparison group and other SGLT-2 inhibitors as the secondary comparison group. | Comparison with other SGLT-2 inhibitors is expected to be underpowered due to the low uptake of SGLT-2 inhibitors other than empagliflozin. |
| | | Multiple | Extending the study | Increasing the study |

| Amendment<br>number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| | | | period until 31 <sup>st</sup> December 2020. | sample size and accounting for the long latency period related to risk of malignancies. |
| | | 9.5 | Updated power calculations. | The power calculations have been updated as a result of extending the study period. |
| | | 9.4.4 | Additional information on potential data sources included. | Additional data sources can be included if the study size will be too small with the current data sources. |
| | | Multiple | Details provided on<br>how fixed-dose<br>combination drugs<br>are processed in the<br>study. | Several fixed-dose<br>combination drugs have<br>become available after<br>the previous protocol<br>version was approved. |

# 5. MILESTONES

| Milestone | Planned Date | Actual date |
|---|---|---|
| Protocol endorsed by the<br>European Medicines Agency<br>(EMA) | Q3 2016 | 19 Sept 2016 |
| Start of data collection | Expected during Q3 2016,<br>depending on final protocol<br>approval by the EMA | 21 Oct 2016 |
| Interim report 24 months | Q1 2017 Will be based on Swedish and the UK data available 24 months after use of empagliflozin is first captured (November 2016) | 13 Mar 2017 |
| Interim report 36 months | Q1 2018 Will be based on Swedish and the UK data available 36 months after use of empagliflozin is first captured (November 2017) | 02 Apr 2018 |
| Interim report 48 months | Q1 2019 Will be based on Swedish and the UK data available 48 months after use of empagliflozin is first captured (November 2018). | 19 Mar 2019 |
| Interim report 60 months | Q1 2020 Will be based on Swedish, the UK and Finnish data available 60 months after use of empagliflozin is first captured (November 2019) | 13 May 2020 |
| Interim report 72 months | Q1 2021 Will be based on Swedish, the UK, and Finnish data available 72 months after use of empagliflozin is first captured (November 2020) | 23 June 2021 |

| Milestone | Planned Date | Actual date |
|---|---|---|
| End of data collection | Q4 2021 Taking into account the database lags, analysis of Swedish and Finnish data through December 2020 will be performed between Q3 2022 and Q3 2023. Analysis of CPRD data through December 2021 will be performed in Q3/Q4 2023. | - |
| Registration in the EU PAS register <sup>1</sup> | Q4 2016 | 30 Nov 2016 |
| Final report of study results | Q2 2024 | - |
| Registration of study results in the EU PAS register | Three months following approval of final study report | - |

Note: Approvals by data protection, data custodian, ethics, and scientific review bodies are pending. Timelines may be impacted by approvals of these bodies, duration of contract reviews, and availability of data and staff at research institutions once contracts and approvals are finalised.

Sponsor to submit to EMA the results of the interim and final study reports within the earliest corresponding PSURs.

<sup>&</sup>lt;sup>1</sup> Website for the EU PAS Register: encepp.eu/encepp\_studies/indexRegister.shtml.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **6.** RATIONALE AND BACKGROUND

Jardiance (empagliflozin), a highly potent and selective inhibitor of the sodium glucose cotransporter 2 (SGLT-2), was approved in Europe in May 2014 for the treatment of type 2 diabetes (T2D) to improve glycaemic control in adults. Synjardy (empagliflozin/metformin hydrochloride) was approved in Europe in May 2015. SGLT-2 is highly expressed in the kidney; as the predominant glucose transporter, it is responsible for the reabsorption of glucose from the glomerular filtrate back into the circulation. Empagliflozin improves glycaemic control in patients with T2D by reducing renal glucose reabsorption [R14-4617].

The recommended starting dose is 10 mg empagliflozin once daily. In patients tolerating empagliflozin 10 mg once daily who have an estimated glomerular filtration rate (eGFR)  $\geq$  60 mL/min/1.73 m2 and need tighter glycaemic control, the dose can be increased to 25 mg once daily. The maximum daily dose is 25 mg [R14-4617].

In Europe, empagliflozin/metformin hydrochloride is available in the following fixed-dose combinations:

- 5 mg empagliflozin plus 850 mg or 1000 mg metformin hydrochloride
- 12.5 mg empagliflozin plus 850 mg or 1000 mg metformin hydrochloride The recommended dose for the fixed-dose combinations is one tablet twice a day [R17-0153]. Currently, little information is available on whether there is a potential increased risk of cancers of the urinary tract associated with empagliflozin use. Clinical data with empagliflozin has not identified or established a potential mechanism for the development of malignancies. However, "urinary tract malignancies" are listed in the Risk Management Plan (RMP) as a potential risk. The inclusion of renal cancer as a potential risk was based on preclinical toxicology findings and clinical cases of bladder cancer observed with other SGLT-2 inhibitors.

As a part of the RMPs for empagliflozin and empagliflozin/metformin hydrochloride agreed upon by the European Medicines Agency (EMA), a post-authorisation safety study (PASS) will be performed to assess the risk of urinary tract malignancies in incident users of empagliflozin, compared to incident users of dipeptidyl peptidase-4 (DPP-4) inhibitors, which is an alternative treatment option to empagliflozin and is prescribed at a similar diabetes progression stage. Prior to the development of the first version of the protocol for this study, a feasibility assessment of three databases in Europe (the CPRD [GOLD and Aurum] and data with potential for linkage (HES and ONS mortality statistics) in the United Kingdom (UK) and the national registers in Sweden and Finland) was performed with the aim to detail the minimum data requirements for the study and to assess, for each potential data source, the data quality, completeness of recorded information for urinary tract malignancies, and possibility of linkage with cancer registries, mortality registries and other data sources. The first version of the protocol included two study countries: Sweden and the UK. with follow-up until 31st December 2019. In version 6.0 of the protocol, the study follow-up was extended until 31st December, 2020 and Finland national registers were included to increase both accumulated patient-years and the number of patients initiating the study drugs.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

In this version of the protocol (Version 7.0), additional steps were taken to increase sample size and follow-up for the UK. CPRD Aurum was added as an additional database to be pooled with CPRD-GOLD and the study period for both CPRD databases was extended to 31st December, 2021.

# 6.1 EPIDEMIOLOGY OF URINARY TRACT MALIGNANCIES IN DIABETES PATIENTS

Based on data from the national cancer registries throughout the Nordic countries, the crude incidence rates (IRs) for urinary tract malignancies (bladder and renal cancers) in the Nordic countries in 2013 was calculated as 43.0 per 100,000 person-years (PY) for the total population and 82.8 per 100,000 PY for individuals over 40 years of age (Table 1) [R15-4873]. As the study population consists of T2D patients who initiate second- or third-line treatment, the majority of the patients are expected to be over 40 years old. The crude incidences of bladder cancer in the UK, as reported through cancer registries to GLOBOCAN, were lower, as compared to the Nordic countries, but rates for renal cancer were comparable (Table 1) [R15-4860]. In both regions, incidences are higher among men.

Table 1 Crude incidence rates per 100,000 person-years for urinary tract cancers, Nordic countries 2013 and the UK 2012

| | <b>Nordic Countries</b> | | | The UK | | |
|---|---|---|---|---|---|---|
| | Male | Female | Total | Male | Female | Total |
| Total Population | | | | | | |
| Bladder | 43.7 | 14.6 | 29.1 | 20.5 | 7.6 | 14 |
| Renal | 17.6 | 10.2 | 13.9 | 19.6 | 11.5 | 15.5 |
| UT (bladder + renal) | 61.3 | 24.9 | 43.0 | 40.1 | 19.1 | 29.5 |
| Age ≥ 40 years | | | | | | |
| Bladder | 87.3 | 27.7 | 56.5 | 47.2 | 16.5 | 31.2 |
| Renal | 34.3 | 18.8 | 26.3 | 44.0 | 23.9 | 33.5 |
| UT (bladder + renal) | 121.6 | 46.5 | 82.8 | 91.3 | 40.4 | 64.7 |

Source: R15-4873; R15-4860

UK=The United Kingdom; UT=Urinary tract

T2D seems to be associated with an increased risk of several types of cancer when compared to the general population. Reviews of recent studies and meta-analyses indicate increased risks for liver, pancreas, colorectal, kidney, bladder, endometrial and breast cancers, as well as non-Hodgkin's lymphoma in patients with T2D [R10-6494, R12-2439, R12-0469]. A population-based cohort study on patients hospitalized with T2D diagnoses in Denmark showed a higher risk of kidney cancers (with the standardized incidence ratios (SIRs) of 1.4 (95% confidence interval (CI); 1.2–1.6) in males and 1.7 (95% CI; 1.4–1.9) in females) and liver cancers (with the SIRs of 4.0 (95% CI; 3.5–4.6) in males and 2.1 (95% CI; 1.6–2.7) in

BI Study Number 1245.97

c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

females) associated with T2D, but not a higher risk for bladder cancer [R15-4869]. Another Swedish inpatient register-based cohort indicated a higher risk of kidney cancer associated with T2D in both women (SIR = 1.7, 95% CI; 1.4-2.0) and men (SIR = 1.3; 95% CI; 1.1-1.6) throughout the duration of follow-up (1-25 years) [R10-6630]. Crude IRs of bladder cancer in patients with T2D range from 38 per 100,000 PY in women from Denmark [R12-1334] to 140-150 per 100,000 PY in men in Sweden and Denmark [R12-0368, R12-1334]. Meta-analyses of observational studies suggest that incidence of kidney cancer in patients with T2D is approximately 40% higher than that in the general population [R13-1812]. The available crude incidence estimates of renal cancer in men with T2D range between 40 and 50 per 100,000 PY in most studies.

Co-existence of hyperinsulinemia and hyperglycaemia in T2D and associated obesity may have a higher associated risk for cancers [R10-6494]. However, there may be additional risks from antidiabetic treatments and insulins, albeit these may be non-significant risks [R10-6494]. Other risk factors of urinary tract cancer are smoking amount and duration ]R15-4868], different occupational and environmental exposures [R15-4865], history of kidney/ureter stones [R15-4863], sex, chronic bladder irritation and infections, genetics and family history, chemotherapy and radiation therapy [R15-4866; R15-4856].

# 6.1.1 Incidence of urinary tract malignancies in the study population in the UK and Sweden observed in the fifth interim report of this study

The country-specific IRs of urinary tract malignancies were estimated in the study population identified in the UK, Sweden and Finland, from 1st August 2014 to 31st December 2020 (2019 for Sweden).

In the UK CPRD GOLD, during a total of 147,020 patient years, 164 urinary tract cancer events were recorded in the study population with an incidence rate of 111.5 (95% CI, 95.7-130.0) per 100,000 patient years. The incidence rate of bladder cancer was 66.7 (95% CI, 54.7-81.2) per 100,000 patient years with a total of 98 events. For renal cancer, the incidence rate was 26.5 (95% CI, 19.4-36.3) per 100,000 patient years with a total of 39 events.

In Sweden, during a total of 210,329 patient years, 346 urinary tract cancer events were recorded in the study population with an incidence rate of 164.5 (95% CI, 148.1-182.8) per 100,000 patient years. The incidence rate of bladder cancer was 104.1 (95% CI, 91.2-118.9) per 100,000 patient years with a total of 219 events. For renal cancer, the incidence rate was 58.0 (95% CI, 48.6-69.3) per 100,000 patient years with a total of 122 events.

In Finland, during a total of 256,947 patient years, 415 urinary tract cancer events were recorded in the study population with an incidence rate of 161.5 (95% CI, 146.7-177.8) per 100,000 patient years. The incidence rate of bladder cancer was 86.8 (95% CI, 76.1-99.0) per 100,000 patient years with a total of 223 events. For renal cancer, the incidence rate was 71.6 (95% CI, 62.0-82.7) per 100,000 patient years with a total of 184 events.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 6.2 EPIDEMIOLOGY OF DIABETES AND DIABETES TREATMENT PATTERNS IN THE UK

The prevalence of diabetes has increased in the UK from 2.8% in 1996 to 4.3% in 2005, and the incidence has increased from 2.7 per 1,000 PY in 1996 to 4.4 per 1,000 PY in 2005. During the period 1996-2005, a change in oral glucose lowering medication use has occurred, predominantly from sulfonylureas to metformin [R11-5320]. Moreover, since 2005-2006, the use of thiazolidinediones has decreased due to concerns about cardiovascular safety, which led to suspension of the rosiglitazone marketing authorisation in the European Union in 2010 [R12-1620]. Together with the introduction in the market of DPP-4 inhibitors, this has changed the selection of second-line treatment regimens, as shown in two studies performed in the UK. One was a cohort study performed in the CPRD from 2000 to 2010, which found that the combination of metformin and DPP-4-inhibitors represented 0.7% of all second-line regimens in 2007, but DPP-4 inhibitors were prescribed in 20.2% of all second-line regimens in 2010 [R14-5249]. On the other hand, the combination of metformin and thiazolidinediones (pioglitazone or rosiglitazone) represented 34% of the all second-line regimens in 2007 but only 9.8% in 2010 [R14-5249]. The other study was performed in The Health Improvement Network (THIN) database, where the annual incidence of prescriptions of thiazolidinediones decreased from 1.2 per 1,000 PY in 2007 to 0.8 per 1,000 PY in 2009, at the same time that "other glucose lowering drugs," including DPP-4 inhibitors, increased from 0.2 per 1,000 PY to 1.1 per 1,000 PY [R14-5244].

As part of the feasibility assessment, patient counts for users of empagliflozin and other glucose lowering medications were extracted from CPRD GOLD database in the UK for the period January 2014 through May 2015 (Table 2). During this time, metformin was the most frequently used glucose lowering medication followed by sulphonylureas, and DPP-4 inhibitors; utilization of empagliflozin was still low.

Table 2 Patient counts by Glucose Lowering Medication category in the UK, Sweden, and Finland

| Drug category | The UK <sup>1</sup> | Sweden <sup>2</sup> | Finland <sup>3</sup> |
|---|---|---|---|
| Biguanides | 149,987 | 235,342 | 246,444 |
| Sulphonylureas | 64,006 | 35,890 | 9,381 |
| Combinations | 2,654 | 2,552 | 39,937 |
| Alpha glucosidase inhibitors | 424 | 703 | None |
| Thiazolidinediones | 9,849 | 1,535 | 4,565 |
| DPP-4 inhibitors | 30,918 | 13,430 | 94,722 |
| Empagliflozin | 108 | 373 | 24,968 |
| Others, excl. insulins | 9,088 | 15,151 | 1,867 |

1 Data from CPRD GOLD, January 2014- July 2015 (end date varies slightly by GP practice). 2 2014. 3 2017

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 6.3 EPIDEMIOLOGY OF DIABETES AND DIABETES TREATMENT PATTERNS IN SWEDEN AND FINLAND

The total age-standardized prevalence of both pharmacologically and non-pharmacologically treated diabetes was 4.69% in 2012 in Sweden. The age-standardized prevalence of pharmacologically treated diabetes increased from 4.19% and 2.99% in 2005/2006 to 5.08% and 3.46% in 2012/2013 in men and women, respectively [R15-4858]. In Finland, 4.3% of women and 7.4% of men aged 45-74 years are diagnosed with diabetes [P19-01624]. In 2016, 5.7% of the Finnish population were dispensed a diabetes drug with a special reimbursement for the costs.

As part of the feasibility assessment, patient counts for users of empagliflozin and other glucose lowering medications were extracted from the Prescribed Drug Register in Sweden for 2014 (<u>Table 2</u>). During this time, metformin was, by far, the most frequently used glucose lowering medication, followed by sulphonylureas and DPP-4 inhibitors; utilization of empagliflozin was still low.

More recent numbers in Finland indicate that metformin was the most frequently used glucose lowering medication in 2016 (Table 2). Empagliflozin use has had a major increase: the number of patients in Finland has increased from 1,007 in 2015 to 24,968 in 2017 [P19-01956].

# 6.4 RISK OF BLADDER CANCER IN PREVIOUS TRIALS OF SGLT-2 INHIBITORS

In a clinical trial comparing empagliflozin with placebo, three (0.1%) and nine (0.4%) cases of bladder cancer were observed in persons exposed to 10 mg and 25 mg empagliflozin, respectively, while five cases (0.2%) were observed among those with exposure to placebo [P19-01957]. Further, dapagliflozin and canagliflozin, in comparison to placebo, did not increase the risk of bladder cancer in clinical trials [R19-2814, P19-07186]. The hazard ratios (HRs) for dapagliflozin, and canagliflozin were 0.57 (95% CI 0.35-0.93) and 0.90 (95% CI 0.47-1.72), respectively. Therefore, contrary to the preclinical toxicology findings, SGLT-2 inhibitors did not show an increased risk of bladder cancer in clinical trials.

### 6.5 RATIONALE FOR THE PROTOCOL AMENDMENT

- 1. The CPRD Aurum database is added to the study data sources. EMA requested to reconsider the inclusion of CPRD Aurum as an additional study database in the UK to capture as many CPRD UK patients as possible, increase the sample size, and improve the study power in this country and in the study overall.
- 2. The study period is extended until 31<sup>st</sup> December, 2021, for CPRD databases (GOLD and Aurum). To increase the sample size and improve study power in the UK, the study period is extended to 31<sup>st</sup> December, 2021, for the CPRD databases.
- 3. Data from the Cancer registry from the United Kingdom (UK) is not included in the study. Data linkage for a sensitivity analysis (Section 8.7.2.3) is not available in time for the final report submission.

## Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1245.97


c03856813-11

- 4. Power calculations are updated using assumptions made from the data available in the 5<sup>th</sup> Interim Report (2021). EMA requested to update the power calculations for the UK considering (1) the inclusion of CPRD Aurum as additional country-specific data source, and (2) using a 1:2 matching ratio for Finland as this matching ratio should be feasible in this country whilst 1:3 will not.
- 5. Additional details regarding the meta-analysis method are included. EMA requested to briefly describe the appropriate methods to combine results obtained from the main analysis performed in the different data sources. This includes describing the meta-analytical techniques such as the meta-analysis model and analysis, describing the handling of heterogeneity, and/or describe the process to identify the most appropriate method for running the meta-analysis.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7. RESEARCH QUESTION AND OBJECTIVES

## **Research Question**

The aim of the study is to assess the risk of urinary tract malignancies in patients initiating empagliflozin compared to patients initiating a DPP-4 inhibitor.

### **Objectives:**

## Primary objectives:

- I. To estimate the adjusted hazard ratios (aHRs) and incidence rates (IRs) of all urinary tract cancers (bladder, renal and other urinary tract cancers) in patients initiating empagliflozin compared to patients initiating a DPP-4 inhibitor
- II. To estimate the aHRs and IRs of bladder cancer in patients initiating empagliflozin compared to patients initiating a DPP-4 inhibitor
- III. To estimate the aHRs and IRs of renal cancer in patients initiating empagliflozin compared to patients initiating a DPP-4 inhibitor

### Secondary objective:

To estimate the aHRs and IR of each primary outcome (all urinary tract cancers, bladder cancer, renal cancer) with respect to:

- a) increasing cumulative dosage of empagliflozin
- b) dosage of empagliflozin prescribed per use (10mg vs 25mg)
- c) time since first dose of empagliflozin



Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 8. RESEARCH METHODS

### 8.1 STUDY DESIGN

This is a non-interventional, comparative, cohort safety study based on European healthcare databases and includes databases from the UK, Sweden and Finland.

The study will use an "incident users" design and compare new users of empagliflozin to new users of DPP-4 inhibitors. The index date will be defined as the date on which each identified new user receives the index prescription for empagliflozin, or a DPP-4 inhibitor. The incident-user design avoids comparing a population predominantly composed of first-time users of a newly marketed drug such as empagliflozin with a population of prevalent users of an older drug who may have stayed on the comparator treatment for a longer time and be less susceptible to the events of interest. To avoid the inclusion of prevalent users, patients will be required to have no exposure to empagliflozin or a DPP-4 inhibitor during the available lookback (pre-index) period [R13-1120, R14-4378].

DPP-4 inhibitors have been selected as the comparator group for several reasons. First, the National Institute for Health and Care Excellence (NICE) appraisal of dapagliflozin (an SGLT-2 inhibitor) recommended that dapagliflozin should be used as described for DPP-4 inhibitors. The NICE Evidence Review Group considered that, overall, "DPP-4 inhibitors are the key comparators for dapagliflozin in both the dual therapy and triple therapy settings" [R13-5134]. Second, DPP-4 inhibitors, SGLT-2 inhibitors, and thiazolidinediones have similar indications and target population, while dual therapy with GLP-1 (glucagon-like peptide-1) analogues has a restricted target population [P14-17374] and metformin and sulfonylureas are typically used earlier in the treatment paradigm. Finally, the use of thiazolidinediones has decreased in recent years, given increasing concerns about their safety (including bladder cancer), and at the same time, use of DPP-4 inhibitors increased, making second-line regimens with DPP-4 inhibitors the most common second-line regimens after metformin with sulfonylurea [R14-5244, R14-5249].

Empagliflozin is usually a second- or third-line treatment for T2D; thus, it is expected that few patients with T2D initiating empagliflozin will be treatment naïve. For the majority of patients, empagliflozin will be added to an existing treatment (e.g., added to metformin), or patients will be switched to empagliflozin (e.g., from metformin plus an oral glucose lowering medication other than the study drugs to metformin plus empagliflozin) due to disease progression, treatment failure, or side effects that may be related to study outcome. Analyses will account for treatment complexity (monotherapy, dual combination therapy, or triple combination therapy) to achieve a fair comparison between groups [R13-1120, R14-4378] and concomitant use of metformin (whether a fixed-dose or free combination). Despite the selection of comparators with similar utilization patterns to empagliflozin, the cohorts created with incident users of DPP-4 inhibitor drug group may have inherent channelling bias wherein the treatment assignment is influenced by a range of factors such as disease progression, comorbidity, treatment history, age, and sex. Additionally, some of these variables lead to increased or decreased risk of cancer. To minimize channelling bias, individuals are matched with similar treatment and clinical history at index date by deriving

BI Study Number 1245.97

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

propensity scores (PS) conditional on factors affecting the treatment and outcome [R13-1120, R14-4378]. Propensity-score-matched cohorts will be derived from the study base by matching patients who initiate empagliflozin with patients who initiate DPP-4 inhibitors at index date with the highest possible matching ratio (1:1, 1:2, or 1:3 using Greedy matching methods). Depending on sample size, combination exposures with metformin will be accounted for through separate PS, stratification, or adjustment. Additional analyses will explore the presence of detection/diagnostic bias as screening for urinary tract signs or symptoms may be more frequently among empagliflozin users. The potential for diagnostic bias will be evaluated and addressed through consideration of the frequency of urine dipstick testing (as captured through albuminuria tests) and stage of cancer at the time of diagnosis (as more early-stage cancers in one group would be suggestive of diagnostic bias).

The primary, secondary, and further analyses utilize a cohort design which will allow direct estimation of the IRs and aHRs of multiple outcomes of interest among new users of empagliflozin compared with new users of a DPP-4 inhibitor. The covariate information will be assessed during the time preceding treatment initiation (varying length look-back (preindex) period) and during follow-up and will include all historical information available for each patient up until occurrence of outcome or censoring (see Section 8.3.3). Follow-up will start 6 months after the index date (12 months in sensitivity analyses) to account for an empirical induction/promotion period (see Section 8.3.5). In the context of data sources such as the CPRD and the Swedish and Finnish national registers, the use of a cohort design has more advantages than limitations compared with the use of a nested case-control (NCC) design—see the appendix discussion in Schneeweiss (2010) [R13-1120] and Patorno et al. (2014) [R14-4378]. Thus, an observational cohort is constructed to study the risk of urinary

The country-level datasets will be analysed separately. Country-level effect size estimates (IRs, aHRs, etc) will be pooled using suitable meta-analysis methods to compute overall estimates.

### 8.2 SETTING

### 8.2.1 Study populations

The source population will include all patients with T2D from the UK, Sweden, and Finland. In the UK, the population will include patients with T2D from the CPRD databases of longitudinal medical records collected from the UK primary care practices (CPRD GOLD and CPRD Aurum). Sensitivity analyses may include a subset of the CPRD GOLD and CPRD Aurum database eligible for linkage to Hospital Episode Statistics (HES) data and/or to Office of National Statistics (ONS) mortality data if linked data with sufficient sample size during the study period are available (see Section 8.4.1). In Sweden and in Finland, patients with T2D in the nationwide registers will be included. All patients with T2D who have purchased at least one prescription of empagliflozin, or a DPP-4 inhibitor during the study
Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

period (2014-2021 for CPRD GOLD and Aurum, 2014-2021 for Sweden and Finland) will be included in the study. Identification of diabetes will be based on medical/prescription records and all non-T2D patients will be excluded.

### 8.2.2 Study period

The study will include individuals who have purchased at least one prescription of empagliflozin, or DPP-4 inhibitors, from 1st August 2014 through 31st December 2020 (31st December 2021 for CPRD). The starting of the study period corresponds to the time of drug licensing (second half of 2014 in all three countries) and subsequent introduction into clinical practice. The number of users in each treatment cohort will be monitored at 24 months after empagliflozin use starts being captured in the data sources (November 2016) and annually thereafter until 2021. The maximum follow-up time for an individual will be seven years for CPRD GOLD and Aurum and 6 years for Sweden and Finland.

### 8.2.3 Index date

The index date will be defined as the date of first purchase/prescription of empagliflozin, or a DPP-4 inhibitor, during the study period (2014-2020).

### 8.2.4 Baseline and look-back (pre-index) period

To characterise the empagliflozin, or DPP-4 inhibitor cohorts at the time of study drug initiation, all information available during the look-back (pre-index) time period will be collected. The look-back time period is defined as the time period ending on the day before the index date. Since all cohort members are required by inclusion criteria to have at least 1 year of data before the index date (baseline period), the look-back period will include at least 365 days during which covariates can be evaluated. For some study participants, data on covariates might be available beyond 1 year prior to the index date; in these cases, all available information will be considered for covariate classification related to diabetes, diabetes medications, and concomitant chronic conditions. For concomitant medications for diseases other than diabetes, the look-back time period will be limited to 180 days prior to the index date.

If the distribution of the duration of look-back time period is different among empagliflozin, or DPP-4 inhibitor categories of look-back time will be created using indicator variables. Those indicator variables will then be used as covariates in the multivariable regression models for outcome prediction, and for PS development, to control for possible differences in availability of information between the empagliflozin and comparator cohorts.

#### 8.2.5 Inclusion and exclusion criteria

The study population will be selected from the broad study population with the following inclusion and exclusion criteria:

#### **Inclusion criteria:**

• Diagnosis of T2D

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- To identify the diagnosis in the UK, lists of codes that have been previously used to identify patients with T2D in the CPRD [P14-16383] will be utilized (Annex 3).
- o For Swedish registers, identification of diabetes will be based on prescription records and the National Diabetes Register; all non-T2D patients will be excluded. The final algorithm to identify patients with T2D in each data source, which might include medication codes and glucose/glycated haemoglobin test results, will be described in the statistical/epidemiological analysis plan (SEAP).
- o In Finnish registers, identification of patients with T2D will be based on prescription records and diagnoses available in various data sources; all non-T2D patients will be excluded. More specifically, all persons with dispensations of empagliflozin, or a DPP-4 inhibitor will be identified. Patients with non-T2D will be identified with the following criteria: special reimbursement of diabetes drugs with an ICD-10 diagnosis for a non-T2D, type 1 diabetes mellitus (T1D), pre-existing T1D before pregnancy, gestational diabetes, malnutrition-related to diabetes mellitus, neonatal diabetes mellitus, other specified diabetes mellitus, diabetes mellitus due to underlying condition, and drug- or chemical-induced diabetes mellitus. The specific diagnosis codes will be included in the SEAP.
- Age over 18 years at index date.
- At least 1 year of membership in the medication database prior to index date; in CPRD, at least 1 year of continuous up-to-standard registration in the CPRD prior to the index date.
  - This is the minimum look-back period and is informative of the history of treatments and other medical conditions in the recent past. Some of the important covariates to be accounted for in matching at index date are derived from the look-back period.

### **Exclusion criteria:**

- Patients with any cancer (excluding non-melanoma skin cancer) recorded at any time prior to the index date (i.e., during the available look-back time).
- Diagnosis of T1D or other specific non-T2D.
- Use of any SGLT-2 inhibitor or any DPP-4 inhibitor (including free and fixed-dose combinations) recorded at any time prior to index date (i.e., during the available look-back time).
- Use of fixed-dose combinations of SGLT-2 inhibitors with DPP-4 inhibitors.
- Diagnosis of or procedures related to end stage renal disease, receipt of renal dialysis recorded, or eGFR ≤15 ml/min at any time prior to index date (i.e., during the available look-back time).

### 8.3 VARIABLES

The final list of variables and operational definitions will be presented in a separate SEAP to be developed prior to the start of data analysis.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8.3.1 Exposures

Empagliflozin (current ATC code A10BK03, previous ATC code A10BX12) is the exposure of interest, free or fixed-dose combination with metformin (ATC code: A10BD20).

The DPP-4 inhibitor comparator exposure group will consist of the following drugs, free or fixed-dose combination with metformin (See Section 8.1 and Annex 4).

- Alogliptin
- Linagliptin
- Saxagliptin
- Sitagliptin
- Vildagliptin

If additional DPP-4 inhibitors are introduced in any of the study countries during the study period, they will also be considered to be members of the corresponding comparator group. Note that use of any of these index drugs prior to index date is an exclusion criterion. Information on whether patients received prior oral glucose lowering therapy or if they were "added on" or "switched to" empagliflozin, or a DPP-4 inhibitor at the time of inclusion in the study will be collected. Patients will be classified according to their treatment complexity as receiving monotherapy, dual combination therapy, or triple combination therapy and according to use of metformin combination therapy (fixed-dose or free combination). (See Section 8.1)

The primary definition of exposure, i.e., as-treated analysis (AT), is defined as an ongoing exposure (free or fixed-dose combination with drugs other than DPP-4 inhibitors and SGLT-2 inhibitors) to one of the following two index drugs or drug groups: empagliflozin or DPP-4 inhibitors (<u>Table 3</u>, Annex 4). Exposure is defined as use of these drugs during the study period starting from 6 months after the index date (see <u>Sections 8.2.3</u> and <u>8.3.5</u>)
As a typical prescription length is one month in the UK and three months in Sweden and Finland, multiple prescriptions are required for a patient to have continuous ongoing treatment at 6 months after index date. Therefore, patients with only one prescription are unlikely to contribute to the AT analysis.

Secondary definitions of exposure include cumulative dosage of empagliflozin use, daily dosage of empagliflozin prescribed per use (10mg vs 25mg), and time since first dose of empagliflozin (Table 3, Annex 4).

Sensitivity analyses of exposure include intention-to-treat (ITT) analyses.

Table 3 Exposure definitions for primary and secondary analyses

| Exposure definition | Description | Time-dependent<br>or Fixed at<br>index date |
|---|---|---|
| Current exposure to study treatment (astreated analysis) | Indicator of current use of empagliflozin, or a DPP-4 inhibitor, either alone or as a combination. | Time-dependent |
| Exposure to Empagliflozin (Intention-to-treat) | Drug purchased/prescribed at index date, which is one of empagliflozin, or a DPP-4 inhibitor. | Fixed at index date |
| Cumulative dosage of empagliflozin use | | |
| Daily dosage of empagliflozin per use | The dosage of empagliflozin prescribed per daily use (10mg vs 25mg). | Time-dependent |
| Time since first dose of empagliflozin Time-dependent cumulative sum of duration since the first use of (exposure to) empagliflozin. | | Time-dependent |
| Treatment complexity | Monotherapy, dual combination therapy, or triple combination therapy (based on predefined groups). | Fixed at index date |
| Switch | Switch from the drug purchased/prescribed on index date to any other drug in the primary exposure. | Time-dependent |
| Concomitant use of insulin | Was empagliflozin an add-on to insulin (yes/no). | Fixed at index date |
| Concomitant use of metformin | Was empagliflozin an add-on to metformin (yes/no). | Fixed at index date |
| Concomitant use of metformin | tived_dose combination or tree | |
| Ever used other oral glucose lowering medication | ucose lowering Use of other oral glucose lowering drugs hased on predefined drug groups in the past | |
| Ever used metformin | Was metformin ever used – taking value 'yes' as soon as one prescription with metformin is purchased. | Time-dependent |

BI Study Number 1245.97

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Exposure definition | Description | Time-dependent<br>or Fixed at<br>index date |
|---|---|---|
| Ever used sulfonylureas | Was sulphonylureas ever used – taking value 'yes' as soon as one prescription with sulphonylureas is purchased. | Time-dependent |
| Ever used thiazolidinediones | Was thiazolidinediones ever used – taking value 'yes' as soon as one prescription with thiazolidinediones is purchased. | Time-dependent |
| Ever used GLP-1 | Was GLP-1 ever used – taking value 'yes' as soon as one prescription with GLP-1 is purchased. | Time-dependent |
| Ever used insulin | Was insulin ever used – taking value 'yes' as soon as one prescription with insulin is purchased. | Time-dependent |

GLP=glucagon-like peptide

### 8.3.2 Outcomes

### 8.3.2.1 Primary outcomes

The outcomes of interest for this study are urinary tract cancers, bladder cancer, and renal cancer. These outcomes will be identified through CPRD GOLD and CPRD Aurum data and the national cancer registries in Sweden and Finland improving confidence in the accuracy and validity of these outcome diagnoses (See Section 8.4).

Date of diagnosis of the first incidence of urinary tract cancers as specified in CPRD GOLD and CPRD Aurum, or in the Swedish or Finnish cancer registry after the entry into the study will be used as the primary outcome date. The urinary tract cancer definition will include malignant neoplasm and carcinoma in situ of the urinary tract. Only the first occurrence of a urinary tract cancer will be captured. Patients with a prior history of cancer, including a prior urinary tract cancer, will be excluded.

In the Swedish and Finnish datasets urinary tract cancer events will be identified from cancer registers using ICD-10 and ICD-O-3 codes (<u>Annex 5</u>). The reporting of all cancer cases is compulsory, and the completeness and quality of the register data are considered good for scientific research [<u>R15-4864</u>, <u>R15-4867</u>, <u>R15-4857</u>, <u>R15-4871</u>].

In CPRD, urinary tract cancer events will be identified in CPRD GOLD and CPRD Aurum using READ and SNOMED codes (Annex 5). A study evaluating the validity of cancer diagnoses in CPRD compared with cancer registry data concluded that recording of cancer diagnoses in the two sources was generally consistent. The predictive value of a CPRD GOLD diagnosis of urinary tract cancer was 92%. Taking all records of cancer in the general

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

practitioner (GP) data, 4% did not occur in the cancer registry data. Differences were generally due to different dates of diagnosis or tumour types [R15-4862].

Sensitivity analyses based on other outcome definitions as well as using a subset of CPRD GOLD and CPRD Aurum with linkage to HES data (Outpatient, HES OP; Admitted Patient Care, HES APC) data, will be performed to address some of the accuracy and validity issues in the primary outcomes (see Section 8.7.2).

### 8.3.3 Covariates

Variables potentially associated with urinary tract cancers, such as socio-demographic variables including age, sex, socioeconomic status, body mass index, smoking and alcohol consumption, laboratory measurements, concomitant medications, comorbidities, and duration of look-back period (see Section 6.1), will be identified for study participants as recorded prior to the index date (see Annex 6 for list of covariates to be included in the study). With the exception of exposure to toxic chemicals such as arsenic, known risk factors for urinary tract cancers are captured in CPRD and the national registers from Sweden and Finland.

Study participants will also be classified by indicator variables on the calendar time of cohort entry (by quarter) whether the index treatment (empagliflozin, or DPP-4 inhibitor) was added to existing medication (adding on), or if the index treatment was initiated as a replacement for another antihyperglycemic medication (switching to empagliflozin, or DPP 4 inhibitor), and whether this treatment was received as monotherapy or as dual or triple combination therapy. A variable indicating whether or not patients were receiving insulin at the index date will also be created.

The confounding due to covariates in this section are to be accounted for at minimum by design or analysis when estimating the risk of urinary tract cancers with the defined

The examples of covariates in Table 4 describe the comorbidities, treatment history, and socio-demographic variables that will considered for inclusion. These variables along with times of occurrence/diagnosis of comorbidities, times of prescription/dispensing of drugs and times of recording of the socio-demographic variables in combination with the exposure and outcome variables define the minimal required dataset.

Table 4

Baseline covariates to be considered for inclusion alternatively or simultaneously in primary, secondary, and further analyses

| | or simulta | neously in p | orimary, seconda | ary, and furt | ner anaryses |
|---|---|---|---|---|---|
| Covariate | Exact<br>matchin<br>g | PS<br>matchin<br>g | Stratificatio<br>n | | |
| Database variable (for CP) | RD only) <sup>1</sup> | | | | |
| Patient database (Aurum vs GOLD) | Yes | Yes | | | |
| Socio-demographic variables | 1 | 1 | | | |
| Age | Yes | Yes | Yes | | |
| Sex | Yes | Yes | Yes | | |
| Socioeconomic status (if available) | | Yes | | | |
| Calendar year of index date | | Yes | | | |
| Duration of look-back period | | Yes | | | |
| Insulin concomitant (or cumulative duration of) use | | Yes | Yes | | |
| Other oral antihyperglycemic medication use | | Yes | | | |
| Comorbidities | | | | | |
| Diabetic complications -<br>diabetic nephropathy-<br>diabetic neuropathy -<br>peripheral vascular<br>diseases - lower limb<br>severity | | Yes | | Yes | Yes |
| Urinary tract-related comorbidities | | Yes | | Yes | Yes |
| Kidney or genitourinary stones | | Yes | | Yes | Yes |

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Covariate | Exact<br>matchin<br>g | PS<br>matchin<br>g | Stratificatio<br>n | Risk set<br>(NCC) /<br>covariat<br>e in<br>MSM <sup>3</sup> | Model<br>adjustmen<br>t <sup>4</sup> |
|---|---|---|---|---|---|
| Prior history of UTI or pyelonephritis | | Yes | | Yes | Yes |
| Liver disease | | Yes | | Yes | Yes |
| eGFR <sup>2</sup> | | Yes | | Yes | Yes |
| Renal impairment | | Yes | | Yes | Yes |
| Prior ICU admission | | Yes | | Yes | Yes |
| Pancreatitis | | Yes | | Yes | Yes |
| BMI (when available) | | Yes | | Yes | Yes |
| Smoking (when available) | | Yes | | Yes | Yes |
| Alcohol use (when available) | | Yes | | Yes | Yes |
| HbA1c (when available) | | Yes | | Yes | Yes |
| Albuminuria testing | | Yes | | Yes | Yes |
| Cardiovascular Diseases (HF, Hypertension, stroke, MI) | | Yes | | Yes | Yes |
| Blood pressure<br>measurements (when<br>available) | | Yes | | Yes | Yes |
| Hypertension | | Yes | | Yes | Yes |
| Stroke | | Yes | | Yes | Yes |
| MI | | Yes | | Yes | Yes |
| Autoimmune disease | | Yes | | Yes | Yes |
| COPD | | Yes | | Yes | Yes |
| Time since first diabetes diagnosis | | Yes | | Yes | Yes |
| Other non-diabetes medications | | | | | |
| Antihypertensives/diureti | | Yes | | | Yes |

| Covariate | Exact<br>matchin<br>g | PS<br>matchin<br>g | Stratificatio<br>n | Risk set<br>(NCC) /<br>covariat<br>e in<br>MSM <sup>3</sup> | Model<br>adjustmen<br>t <sup>4</sup> |
|---|---|---|---|---|---|
| cs | | | | | |
| Non-steroidal anti-<br>inflammatory drugs<br>(NSAIDs) | | Yes | | | Yes |
| Oral steroids | | Yes | | | Yes |
| Statins, fibrates | | Yes | | | Yes |
| Lipid modifying agents | | Yes | | | Yes |
| Zoledronic acid | | Yes | | | Yes |
| Antibiotics | | Yes | | | Yes |

- 1 This variable will be present only for CPRD data. It will indicate which database (GOLD or Aurum) the patient data was extracted from-
- 2 Time-dependent eGFR estimate will be computed with the CKD-Epi equation from serum creatinine measurements, where available.
- 3 Sensitivity analyses
- 4 Covariates considered for inclusion if not balanced after PS matching

BMI=body mass index; COPD=chronic obstructive pulmonary disease; eGFR=estimated glomerular filtration rate; HbA1c=glycated haemoglobin A1c; HF=heart failure; ICU=intensive care unit; MI=myocardial infarction; MSM=marginal structural model; NCC=nested case-control; PS=propensity score; UK CPRD=The United Kingdom Clinical Practice Research Datalink; UTI=urinary tract infection.

### 8.3.4 Censoring of follow-up time

The following events lead to censoring: all-cause mortality, emigration, patient transfer, meeting specific exclusion criteria (see exclusion criteria in Section 8.2.5) and end of study period. Follow-up times will be censored at any of these events, whichever occurs first. In the primary AT analysis discontinuation of index drug treatment is an additional censoring variable. Treatment discontinuation is defined either by

- A switch from the index drug to any other drugs (empagliflozin, DPP-4 inhibitor, or other SGLT-2 inhibitor), or to a fixed-dose combination of a SGLT-2 inhibitor with a DPP-4 inhibitor (identified from the ATC class A10BD) plus a 3-month period following the switch, or
- As the stop date plus a 3-month period following it. The stop date is the end date of the first continuous exposure period of the index drug, where continuous treatment is defined as having consecutive prescriptions separated by 30 days or less (Figure 1).

The 3-month period after the switch or the stop date is used to allow for a delay in the diagnosis of cancer [R16-2539]. In a sensitivity analysis this time period is extended to 6 months.

# Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1245.97


c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Switch to a fixed-dose combination including the same index drug and drugs other than DPP-4 inhibitors and SGLT-2 inhibitors is not considered a censoring variable (for example, switch from sitagliptin to a fixed-dose combination including sitagliptin and pioglitazone).



Figure 1 Discontinuation of index drug due to stopping of index drug or switching of index drug. In the primary analysis follow-up is censored at treatment discontinuation.

### 8.3.5 Follow-up time

For the primary AT analyses, the follow-up time (time at risk) will begin 6 months after the index date (lag period to account for empirical induction/promotion period of cancer) and end at urinary tract (bladder, renal or other) cancer or at any of the censoring events including discontinuation of index drug treatment.

For the sensitivity ITT analyses, the follow-up time will begin 6 months after the index date and end at urinary tract (bladder, renal or other) cancer or any of the censoring events excluding treatment discontinuation of index drug.

Patients with censored follow-up time will not be able to re-enter study cohort at a later time point. Follow-up will not be censored if oral or injectable glucose lowering drugs other than the index drugs are prescribed in addition to empagliflozin, a DPP-4 inhibitor, or a SGLT-2 inhibitor after the index date.

The lag period of 6 months is to account for an empirical induction/promotion period. Information in the first 6 months after the index date (i.e., first 6 months of follow-up) will be excluded, including patients with less than 6 months of follow-up and all occurrences of cancer within the first 6 months of follow-up, in order to consider a biologically meaningful induction/promotion time window. Sensitivity analyses will expand the lag period to 12 months.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8.4 DATA SOURCES

Prior to the development of the protocol for this study, a feasibility assessment of three databases in Europe (CPRD [GOLD and Aurum] and data with potential for linkage [HES (Outpatient and Admitted Patient Care), and ONS mortality statistics] in the UK and the national registers in Sweden and Finland) was performed with the aim to detail the minimum data requirements for the study and to assess, for each potential data source, the data quality, completeness of recorded information for urinary tract malignancies, and possibility of linkage with cancer registries, mortality registries and other data sources. The minimal data requirements for data sources which were assessed are listed in Table 5.

Table 5 Minimum data requirements and data availability for the UK and the national registries in Sweden and Finland.

| | The UK | | | Swed | Sweden | | | Finland | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | CPRD (GOLD and Aurum) | HES | Mortal<br>ity | Patient | Prescri<br>ption | Cancer | Cause<br>of | <b>Diabet</b> es | НІГМ<br>О | AvoHI<br>LMO | Special<br>Reimb | Prescip<br>tions | Cause<br>of | Cancer<br>s | EMR<br>databa |
| Age | X | X | X | X | X | X | X | X | X | X | - | X | X | X | X |
| Sex | X | X | X | X | X | X | X | X | X | X | - | X | X | X | X |
| Medication | X | - | | $x^3$ | X | - | - | <b>x</b> <sup>5</sup> | - | - | - | X | - | X | - |
| DDD | X | - | - | X | X | - | - | - | - | - | - | X | - | - | - |
| Purchase date | $\mathbf{x}^1$ | - | - | X | X | - | - | - | - | ı | - | X | - | ı | - |
| Diagnoses | X | X | - | x <sup>4</sup> | - | X | - | X | X | X | $\mathbf{x}^7$ | x <sup>9</sup> | - | X | - |
| Date of diagnosis | X | x | 1 | X | - | X | - | - | X | X | <b>x</b> <sup>8</sup> | - | - | X | - |
| Time of death | - | - | X | ı | - | X | X | - | - | ı | - | - | X | X | - |
| Cause of death | - | - | X | - | - | X | X | - | - | ı | - | - | X | X | - |
| Smoking | X | - | - | - | - | - | - | X | x <sup>6</sup> | <b>x</b> <sup>6</sup> | - | - | - | - | X |
| BMI | X | - | - | - | - | - | - | X | x <sup>6</sup> | x <sup>6</sup> | - | - | - | - | X |
| HbA1c | X | - | - | - | - | - | - | X | - | - | - | - | - | - | X |

x = available in the register, - = not available in the register

## Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1245.97


c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 1 Prescription date; 2 Month and year; 3 Treatment given in hospitals (no full coverage); 4 No primary care data; 5 Only type of medication; 6 Partial availability based on applicable diagnosis codes; 7 Only chronic diseases included in the special reimbursement scheme; 8 Start and end dates of the special reimbursement; 9 In case a special reimbursement was included in the purchase
- AvoHILMO=Register of primary health care visits, BMI=body mass index, CPRD=Clinical Practice Research Datalink, DDD=Defined daily dose, EMR=electronic medical record, HbA1c=Glycated haemoglobin A1c, HES=Hospital Episode Statistics (Outpatient data, and Admitted Patient Care data), HILMO=Care register for health care; UK =The United Kingdom

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8.4.1 The United Kingdom Clinical Practice Research Datalink (CPRD)

The UK CPRD data contains the anonymised longitudinal medical records managed by GPs working in the National Health Service (NHS) primary care setting. The data contains demographic information, diagnoses, prescriptions, tests and referrals. This study will use data extracted from CPRD GOLD [R16-1231] and CPRD Aurum [R19-1534].

### **CPRD GOLD**

CPRD GOLD data [R16-1231] cover approximately 8.8% of the UK population, including practices in England, Wales, Scotland and Northern Ireland. Data has been collected prospectively since 1987. Approximately 54% of CPRD GOLD practices take part in the English linkage program (CPRD GOLD-HES subset), which includes patient-level linkage to the inpatient data (HES), allowing for hospitalization diagnoses and procedures to be captured [R19-2928]. Records in both settings include the unique NHS number, which is used for linkage purposes. In a similar way, CPRD GOLD data is linked to the UK mortality data (including date and cause of death). Protocols using CPRD GOLD and linked data are subject to approval by an Independent Scientific Advisory Committee.

#### CPRD Aurum

CPRD Aurum was established in October 2017 [R19-1534], and therefore, its feasibility could not be assessed before starting the present study.

CPRD Aurum data cover approximately 13% of the population in England (as of September 2018) [R19-1534]; however, recruitment of additional practices is ongoing. Similar to CPRD GOLD, the data available in CPRD Aurum can be linked with other data sources using the NHS number. In total, 93% of the participating practices take part in the linkage program (R19-2928). The same variables are available in CPRD GOLD and in CPRD Aurum.

The main difference between CPRD Aurum and CPRD GOLD is that the data has been recorded from different practices using different software [R19-1534]. As practices migrate from one software to the other, they will also migrate from the GOLD database to the Aurum database. Duplicate historical data will then be available for patients from these practices in both GOLD and Aurum. This possibility will be taken into account as both CPRD GOLD and CPRD Aurum data are incorporated in this study. The data holder (CPRD) will provide a list of migrated (GOLD to Aurum) practices. As Aurum will provide the longest follow-up, the data of patients from migrating practices present in both databases will be removed from the GOLD data but retained in the Aurum data.

### Linkage

Based on the feasibility assessment before this study, the UK data sources evaluated (CPRD GOLD and data with potential for linkage - HES, ONS mortality statistics) met the minimal data requirements (Table 5). Similar results were expected for the CPRD Aurum. The following UK data sources are considered for linkage with CPRD: HES (Outpatient data and Admitted Patient Care data), and Office for National Statistics (ONS) mortality sources. In the UK, the full study data including follow-up period until the end of 2021, will be available

# Protocol for non-interventional studies based on existing data BI Study Number 1245.97

c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

in March 2022. The primary analyses will be based on CPRD GOLD and CPRD Aurum data; sensitivity analyses may include linked HES (Outpatient and Admitted Patient Care data) and ONS data, if linked data with sufficient sample size during the study period are available (Section 8.7.2.3.3).

To determine renal impairment, eGFR values will be extracted from CPRD. Additionally, information on important covariates such as proxies of socioeconomic position, number of albuminuria tests, blood pressure measurements will be extracted.

### 8.4.2 Swedish national registries

Sweden has a well-developed population-wide register system with longitudinal follow-up data. The persons are identified in the registers with a unique personal identification number (PID) and thus the records can be linked for research purposes on subject level between the registers. Permissions to use the data may be received upon providing a research plan to the authorities responsible for the registers. The protocol is also subjected to relevant Ethical Committee's review and approval. The data permit processes and timelines for data permit granting by the authorities responsible for the registers vary between different registers and countries, as well as the requirements for the local research collaboration and the publication of results [R15-4861].

The nationwide prescription register contains information on outpatient medication purchases in pharmacies. All prescribed medicines purchased in community pharmacies are included irrespective of reimbursement status.

Based on the feasibility assessment, the Sweden national registers met the minimal data requirements (<u>Table 5</u>). The following data sources will be used to construct the Sweden cohort by linkage: The National Patient Register, the Swedish Prescribed Drug Register, the Swedish Cancer Register, the Causes of Death Register, the National Diabetes Register, and the Longitudinal integration database for health insurance and labour market studies.

To determine renal impairment, eGFR values will be extracted from the National Diabetes Register. Information on important covariates such as number of albuminuria tests and blood pressure measurements will also be extracted from the National Diabetes Register. Further, proxies of socioeconomic position will be obtained from the Longitudinal integration database for health insurance and labour market studies.

The study data will be extracted from the relevant registers using the following general process. First, patients in the study cohort with the unique PID number are identified from the prescription register. A unique dummy study identification number (SID) is created for each PID by the prescription register holder. The list with the PID-SID pairs will be provided from the prescription register holders to the other register holders. Each register holder extracts the relevant data according to the study protocol and links the data to the PID-SID list. Subsequently, the register holders decode the data by destroying the key between the PID and SID permanently and provides the de-identified study data to the applicant. Thus, only de-identified data will be provided for performing the analysis of the study data. In Sweden, the full study data including follow-up period until the end of 2020 will be available during in March 2022.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8.4.3 Finnish data sources

BI Study Number 1245.97

An additional, feasible data source in Europe includes the national registers in Finland, which were evaluated in the feasibility assessment before this study.

As in Sweden, Finland has a well-developed population-wide register system with longitudinal follow-up data. The persons are identified in the registers with a unique PID and thus the records can be linked for research purposes on subject level between the registers. Further, the data obtained from registers can be linked with data obtained from the EMR databases.

The following Finnish nationwide data sources will be included: Care register for health care (HILMO), Register of primary health care visits (AvoHILMO), Special reimbursement register, Prescription register, Cause of death register, Cancer register, Population register centre, and Statistics Finland (Table 5). HILMO and AvoHILMO include diagnoses associated with healthcare encounters in specialized and primary care, respectively. The Special reimbursement register will be used for identification of chronic comorbidities. This register includes patients who are entitled for special refunds of medicine expenses based on their chronic conditions. The Finnish nationwide Prescription register contains information on outpatient medication purchases in pharmacies. The register contains information on all purchased prescribed medicines within the reimbursement scheme. Cause of death register includes time of death and the cause of death classified according to the ICD categorization. Cancer register includes information on all diagnosed cancers, details of the tumour, and description of treatment.

The study data will be extracted from these registers using the general process as described above for Sweden (Section 8.4.2). Information about highest level of education will be obtained as a proxy for socioeconomic status from Statistics Finland, and information on patient's place of residence and migration will be obtained from Population register centre.

Further, to obtain data on important potential confounders, specifically BMI, blood pressure, smoking, and laboratory measures such as HbA1c and eGFR, EMR databases will also be included in the study. Four regional EMR databases (Helsinki, Espoo, Vantaa, and Helsinki University Hospital [HUS] area), covering both primary and secondary care in the capital area of Finland, will be contacted separately to obtain access to their data. The data obtained from different data sources will be linked as described previously (Section 8.4.2).

Permissions to use the data may be received upon providing a research plan to the authorities responsible for the registers. The protocol is also subjected to relevant Ethical Committee's review and approval. The data permit processes and timelines for data permit granting by the authorities responsible for the registers vary between different registers and countries, as well as the requirements for the local research collaboration and the publication of results [R15-4861].

In Finland, all the data will be delivered to and analysed in the remote access server environment provided by the national permit authority Findata. The data holders will extract the relevant data and deliver it to Findata for pseudonymization. Before data delivery to the

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Findata server environment, the data holders will collect and manage data according to their own standards. After the data is delivered to the Findata server environment by the data holders, will process the data.

will use the study identification numbers for data linkage on individual level. will have access to pseudonymized raw data without PINs. Therefore, the researchers at identified.

In Finland, the full study data including follow-up period until the end of 2020 will be available in June 2022.

### 8.4.4 Additional potential data sources

Beside the data sources evaluated originally in the UK, Sweden, and Finland, none of the holders of other databases have been contacted for participation in the study so far, and further feasibility assessments are required to insure the validity of urinary cancer case identification. It is important for the choice of the appropriate data source to have the appropriate information on cancer and important risk factors included.

Potential additional data sources for this study have been assessed (Annex 1). In addition to those described above, Danish nationwide registers, PHARMO Database Network (Netherlands), Spanish regional registers, and Maccabi Healthcare Services database (Israel) are feasible for inclusion in the study.

### 8.5 STUDY SIZE

The study size will be driven by the uptake of empagliflozin and the primary comparator (DPP-4 inhibitors) in the UK, Sweden, and Finland. Originally, it was expected that by the end of 2019, approximately 18,000 empagliflozin-treated patients will accumulate in the CPRD and Swedish databases. However, based on the conservative estimates from the fifth interim analysis (Annex 1), the expected sample size is higher than anticipated. Taking into account the addition of Finland, the addition of CPRD Aurum, and the extension of the study period (end of 2020 for Sweden and Finland, end of 2021 for CPRD), a total of approximately 67,490 empagliflozin users are expected to be eligible for inclusion in the study (Table 6). However, the number of patients available for analysis may be lower. Given the observed patient numbers, it is expected that the maximum achievable matching ratios will be 1:3 for UK CPRD (GOLD and Aurum), 1:1 for Sweden, and 1:2 for Finland.

Table 6

Observed and expected number of patients eligible for inclusion in the study population, by study drug group (including fixed-dose combinations with metformin), by study country and overall, using an arithmetic growth assumption.

| Year | Study drug group | Finland | Sweden | CPRD GOLD | CPRD<br>Aurum4 | Pooled |
|---|---|---|---|---|---|---|
| | Empagliflozin | 0 | 0 | 5 | | 5 |
| 2014 <sup>1</sup> | DPP 4-inhibitors | 5,824 | 3,214 | 2,555 | | 11,593 |
| | Other SGLT-2 inhibitors | 127 | 662 | 683 | | 1,472 |
| | Empagliflozin | 91 | 629 | 157 | | 877 |
| 2015 <sup>1</sup> | DPP 4-inhibitors | 14,130 | 10,305 | 6,851 | | 31,286 |
| | Other SGLT-2 inhibitors | 320 | 1,537 | 2,065 | | 3,922 |
| | Empagliflozin | 2,201 | 2,181 | 897 | | 5,279 |
| 2016 <sup>1</sup> | DPP 4-inhibitors | 11,391 | 12,126 | 5,648 | | 29,165 |
| | Other SGLT-2 inhibitors | 1,463 | 1,183 | 1,740 | | 4,386 |
| | Empagliflozin | 3,725 | 4,811 | 1,391 | | 9,927 |
| 20171 | DPP 4-inhibitors | 7,402 | 13,677 | 4,577 | | 25,656 |
| | Other SGLT-2 inhibitors | 1,475 | 1,191 | 1,493 | | 4,159 |
| | Empagliflozin | 4,293 | 8,738 | 1,536 | | 14,567 |
| 2018 <sup>1</sup> | DPP 4-inhibitors | 6,959 | 12,798 | 4,158 | | 23,915 |
| | Other SGLT-2 inhibitors | 1,610 | 1,030 | 1,470 | | 4,110 |
| | Empagliflozin | 5,182 | 10169 | 1,846 | | 17,197 |
| 2019 <sup>1</sup> | DPP 4-inhibitors | 6,158 | 11,673 | 3,622 | | 21,453 |
| | Other SGLT-2 inhibitors | 1,853 | 1,061 | 1,665 | | 4,579 |
| | Empagliflozin | 2,777 | 5,806 | 1,541 | | 10,124 |
| $2020^{2}$ | DPP 4-inhibitors | 2,215 | 4,688 | 2,210 | | 9,113 |
| | Other SGLT-2 inhibitors | 1,201 | 653 | 1,369 | | 3,223 |
| | Empagliflozin | | | 969 | | |
| 2021 <sup>3</sup> | DPP 4-inhibitors | | | 1,051 | | |
| | Other SGLT-2 inhibitors | | | 726 | | |
| Та4-1 | Empagliflozin | 18,269 | 32,334 | 8,342 | 8,545 | 67,490 |
| Total | DPP 4-inhibitors | 54,079 | 68,481 | 30,672 | 59,283 | 212,515 |

# Protocol for non-interventional studies based on existing data BI Study Number 1245.97

c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Year | Study drug group | Finland | Sweden | CPRD GOLD | CPRD<br>Aurum4 | Pooled |
|---|---|---|---|---|---|---|
| | Other SGLT-2 inhibitors | 8,049 | 7,317 | 11,211 | 25,277 | 51,854 |

- 1 Observed number of patients.
- 2 Observed number of patients until 30th June for Sweden and Finland and until 31st December for UK CPRD GOLD, taking into account the extension of the study period to the end of 2021 for UK CPRD.
- 3 Expected number of patients (arithmetic growth assumption given observed numbers in previous years) between 1st January and 30th June, taking into account the 6 months minimum follow-up.
- 4 Only aggregate level data up (2014-2020) of was available for CPRD Aurum. Patient numbers were extrapolated based on assumptions derived from CPRD GOLD data, taking into account the extension of the study period to the end of 2021 DPP-4=dipeptidyl peptidase-4 inhibitors; SGLT-2=sodium glucose co-transporter-2 inhibitors; UK=the United Kingdom

The power to detect relative risks of 1.5 and 2 was determined for each of the study outcomes for each individual country (Table 7) and for the final random-effects meta-analysis (Table 8). For the single-country analyses, power computations were based on HRs derived from Cox models. For the meta-analysis, simulations were used to estimate country-level HRs which were then entered into random-effects meta-analysis models as described in Section 8.7.1.4. All power computations were based on the expected number of individuals exposed to empagliflozin eligible for inclusion in the study and the observed country-level IRs of urinary tract cancers, bladder cancer and renal cancer in the study population as reported in the 5th Interim Report. The expected averages of follow-up time were 2.4 years for UK CPRD, 2.2 for Sweden, and 2.4 for Finland, as reported in the 5th Interim Report. Matching ratios of empagliflozin initiators to initiators of DPP-4 inhibitors were fixed at 1:3 for UK CPRD, 1:1 for Sweden, and 1:2 for Finland. These are the highest achievable matching ratios given expected patient numbers. For computing the meta-analysis power, these assumptions were used to simulate for each country separately individual level time-to-event data from each drug cohort following an exponential distribution given the expected number of empagliflozin initiators, the expected matching ratio, the observed incidence rates as the baseline rate in the DPP-4 cohort. The hazard ratio for each simulation run was determined by drawing from a normal distribution with a mean of the natural logarithm of the target hazard ratio (1.5 or 2.0) and a standard deviation of 0.1. These individual time-to-event data were then entered into a Cox proportional hazard model for each country to compute a simulated hazard ratio. For each simulation, the country-level hazard ratios were entered into a random-effects meta-analysis level, and the resulting p-value of the pooled estimate was retained. Simulations were run 500 times and power was computed as the proportion of simulations for which the p-value of the pooled estimate was inferior to 0.5. The power calculations show that anticipated study sample size would ensure sufficient power at the meta-analysis level to detect the targeted effect size of < 1.6 for urinary tract cancers and bladder cancer and the targeted effect size of < 2.0 for renal cancer, with at least 80% power and a type 1 error probability of 5% under the expected matching ratios. Power at the meta-analysis level to detect an effect size of 1.5 is expected to be of 93.6% for urinary tract cancer and 84.0% for bladder cancer. Power at the meta-analysis level to detect an effect size of 2.0 is expected to be of 97.0% for renal cancer.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7

Power for different effect sizes for single-country analyses based on Cox models with a type 1 error probability of 5%, given country-level observed incidence rates, expected numbers of empagliflozin initiators, expected follow-ups, and expected matching ratios.

| Effect size<br>(Hazard ratio) | Urinary tract cancer | Bladder<br>cancer | Renal cancer |
|---|---|---|---|
| UK CPRD <sup>1</sup> | , | | |
| 1.5 | 63.7% | 43.1% | 20.3% |
| 2.0 | 99.1% | 91.7% | 55.9% |
| Sweden <sup>2</sup> | | | • |
| 1.5 | 85.1% | 66.6% | 42.9% |
| 2.0 | >99.9% | 99.0% | 89.4% |
| Finland <sup>3</sup> | | | • |
| 1.5 | 80.6% | 54.3% | 46.7% |
| 2.0 | 99.9% | 96.8% | 93.4% |

<sup>1</sup> Includes both CPRD GOLD and Aurum; Observed IRs of 111.5, 66,7, and 26.5 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected follow-up of 2.4, matching ratio of 1:3, and expected number of empagliflozin initiators of 16,360.

UK CPRD=The United Kingdom Clinical Practice Research Datalink

Table 8

Power of meta-analyses for a type 1 error probability of 5% for different effect sizes, given country-level observed incidence rates, expected number of empagliflozin initiators, expected average follow-ups, and expected matching ratios.

| Effect size<br>(Relative risk /<br>hazard ratio) | Urinary tract cancer | Bladder cancer | Renal cancer |
|---|---|---|---|
| 1.5 | 93.6% | 84.0% | 68.2% |
| 2.0 | >99.9% | 99.6% | 97.0% |

For UK CPRD (GOLD and Aurum): observed IRs of 111.5, 66,7, and 26.5 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected follow-up of 2.4, matching ratio of 1:3, and expected number of empagliflozin initiators of 16,360.

For Sweden: observed IRs of 164.5, 104.1, and 58.0 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected follow-up of 2.2, matching ratio of 1:1, and expected number of empagliflozin initiators of 32,334.

<sup>2</sup> Observed IRs of 164.5, 104.1, and 58.0 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected follow-up of 2.2, matching ratio of 1:1, and expected number of empagliflozin initiators of 32,334.

<sup>3</sup> Observed IRs of 161.5, 86.8, and 71.6 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected follow-up of 2.4, matching ratio of 1:2, and expected number of empagliflozin initiators of 18,269.

BI Study Number 1245.97

### c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For Finland: observed IRs of 161.5, 86.8, and 71.6 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected follow-up of 2.4, matching ratio of 1:2, and expected number of empagliflozin initiators of 18,269.

The minimum detectable effect sizes for each outcome were computed given the observed and expected IRs, average follow-ups, matching ratios, and number of empagliflozin initiators for single-country analyses as well as for a random-effects meta-analysis (Table 9). At the meta-analysis level, the minimum detectable effect sizes were 1.37 for urinary tract cancers, 1.47 for bladder cancer, and 1.62 for renal cancer.

Table 9

Minimum detectable effect sizes (Hazard Ratios) given country-level observed incidence rate, expected sample sizes, expected average follow-ups, and matching ratios for single-country analyses and meta-analyses for a type 1 error probability of 5%.

| | Urinary tract cancer | Bladder cancer | Renal cancer |
|----------------------|----------------------|----------------|--------------|
| UK CPRD <sup>1</sup> | 1.62 | 1.82 | 2.40 |
| Sweden <sup>2</sup> | 1.46 | 1.60 | 1.85 |
| Finland <sup>3</sup> | 1.50 | 1.70 | 1.78 |
| Meta-analysis | 1.37 | 1.47 | 1.62 |

<sup>1</sup> Includes both CPRD GOLD and Aurum; Observed IRs of 111.5, 66,7, and 26.5 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected follow-up of 2.4, expected number of empagliflozin initiators of 16,360, and matching ratio of 1:3.

The study sizes for each individual country required to detect a relative risk of 1.5 and 2.0, with 80% power under the expected country-level matching ratios and observed country-level IRs were computed for each study country individually (Table 10) and for a random-effects meta-analysis (<u>Table 11</u>). At the meta-analysis level, the required country-level sample sizes to detect an effect size of 1.5 for urinary tract cancer are 9,076, 17,377, and 9,818 for UK CPRD, Sweden, and Finland, respectively. For detecting an effect size of 2.0 for renal cancer at the meta-analysis level, the required sample sizes are 6,534, 12,510, and 7,069 for UK CPRD, Sweden, and Finland, respectively.

<sup>2</sup> Observed IRs of 164.5, 104.1, and 58.0 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected follow-up of 2.2, expected number of empagliflozin initiators of 32,334, and matching ratio of 1:1.

<sup>3</sup> Observed IRs of 161.5, 86.8, and 71.6 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected follow-up of 2.4, expected number of empagliflozin initiators of 18,269, and matching ratio of 1:2. UK CPRD=The United Kingdom Clinical Practice Research Datalink

Table 10

Required sample sizes in each study country to estimate different effect sizes for the three primary endpoints in the single-country analyses with at least 80% power and a type 1 error probability of 5%, given country-level incidence rates, expected average follow-ups, and expected matching ratios.

| | HR=1.5 | | | HR=2 | | |
|---|---|---|---|---|---|---|
| Primary endpoints | UK<br>CPRD <sup>1</sup><br>(1:3) | Sweden <sup>2</sup> (1:1) | Finland <sup>3</sup> (1:2) | UK<br>CPRD <sup>1</sup><br>(1:3) | Sweden <sup>2</sup> (1:1) | Finland <sup>3</sup> (1:2) |
| All Urinary tract cancers | 25,810 | 28,151 | 17,999 | 7,072 | 8,665 | 5,276 |
| Bladder<br>cancer | 41,550 | 44,523 | 33,543 | 11,846 | 13,707 | 9,835 |
| Renal cancer | 104,474 | 79,991 | 40,665 | 29,788 | 24,630 | 11,924 |

<sup>1</sup> Includes both CPRD GOLD and Aurum; Observed IRs of 111.5, 66,7, and 26.5 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively and expected follow-up of 2.4.

HR=Hazard ratio; UK CPRD=The United Kingdom Clinical Practice Research Datalink

<sup>2</sup> Observed IRs of 164.5, 104.1, and 58.0 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively expected follow-up of 2.2.

<sup>3</sup> Observed IRs of 161.5, 86.8, and 71.6 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively expected follow-up of 2.4.

Table 11

Required sample sizes in each study country to estimate different effect sizes for the three primary endpoints in the meta- analyses with at least 80% power and a type 1 error probability of 5%, given country-level incidence rates, expected average follow-ups, and expected matching ratios.

| | HR=1.5 | | | HR=2.0 | | |
|---|---|---|---|---|---|---|
| Primary endpoints | UK<br>CPRD <sup>1</sup><br>(1:3) | Sweden <sup>2</sup> (1:1) | Finland <sup>3</sup> (1:2) | UK<br>CPRD <sup>1</sup><br>(1:3) | Sweden <sup>2</sup> (1:1) | Finland <sup>3</sup> (1:2) |
| All Urinary tract cancers | 9,076 | 9,076 | 9,076 | 2,561 | 4,903 | 2,770 |
| Bladder<br>cancer | 15,505 | 29,687 | 16,773 | 4,058 | 7,769 | 4,390 |
| Renal cancer | 25,252 | 48,350 | 27,318 | 6,534 | 6,534 | 6,534 |

<sup>1</sup> Includes both CPRD GOLD and Aurum; Observed IRs of 111.5, 66,7, and 26.5 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively and expected follow-up of 2.4.

HR=Hazard ratio; UK CPRD=The United Kingdom Clinical Practice Research Datalink

The average follow-up time required to achieve 80% power to detect HRs of 1.5 and 2.0 with the expected number of patients (<u>Table 6</u>) and observed IRs was evaluated for each of the study outcomes for the country-level analyses (<u>Table 12</u>) and for a random-effects meta-analysis (<u>Table 13</u>).

<sup>2</sup> Observed IRs of 164.5, 104.1, and 58.0 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively expected follow-up of 2.2.

<sup>3</sup> Observed IRs of 161.5, 86.8, and 71.6 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively expected follow-up of 2.4.

Table 12

Required follow-up time (years) to achieve 80% power in country-level analyses with a type 1 error probability of 5% for different effect sizes for the three primary endpoints given country-level observed incidence rates, expected sample sizes, and expected matching ratios

| Matching | Hazard ratio | Urinary tract cancer | Bladder cancer | Renal cancer |
|---|---|---|---|---|
| UK CPRD¹ | | | | |
| 1:3 | 1.5 | 3.03 | 4.73 | 11.13 |
| | 2.0 | 1.22 | 1.71 | 3.54 |
| Sweden <sup>2</sup> | | | | |
| 1:1 | 1.5 | 1.99 | 2.86 | 4.73 |
| | 2.0 | 0.96 | 1.23 | 1.81 |
| Finland <sup>3</sup> | | | | |
| 1:2 | 1.5 | 2.38 | 4.00 | 4.75 |
| | 2.0 | 1.05 | 1.53 | 1.75 |

<sup>1</sup> Includes both CPRD GOLD and Aurum; Observed IRs of 111.5, 66,7, and 26.5 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected number of empagliflozin initiators of 16,360, and matching ratio of 1:3.

<sup>2</sup> Observed IRs of 164.5, 104.1, and 58.0 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected number of empagliflozin initiators of 32,334, and matching ratio of 1:1.

<sup>3</sup> Observed IRs of 161.5, 86.8, and 71.6 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected number of empagliflozin initiators of 18,269, and matching ratio of 1:2.

UK CPRD=The United Kingdom Clinical Practice Research Datalink

Table 13

Required follow-up time (years) in each study country to achieve 80% power for the meta-analysis with a type 1 error probability of 5% for different effect sizes for the three primary endpoints given country-level observed incidence rates, expected sample sizes, and expected matching ratio

| Matching | Hazard ratio | Urinary tract cancer | Bladder cancer | Renal cancer |
|---|---|---|---|---|
| UK CPRD¹ | | | | |
| 1:3 | 1.5 | 1.38 | 2.05 | 3.08 |
| | 2.0 | 0.74 | 0.91 | 1.20 |
| Sweden <sup>2</sup> | | | | |
| 1:1 | 1.5 | 1.38 | 2.04 | 3.07 |
| | 2.0 | 0.74 | 0.91 | 1.20 |
| Finland <sup>3</sup> | | | | |
| 1:2 | 1.5 | 1.50 | 2.22 | 3.35 |
| | 2.0 | 0.81 | 0.99 | 1.31 |

<sup>1</sup> Includes both CPRD GOLD and Aurum; Observed IRs of 111.5, 66,7, and 26.5 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected number of empagliflozin initiators of 16,360, and matching ratio of 1:3.

Based on the feasibility assessment before this study and the interim reports, utilization of empagliflozin in the UK and Sweden is still low. Accrual of empagliflozin users is monitored in the data sources as described in Section 8.7.1.7. The number of users in each treatment cohort has been monitored at 24 months after empagliflozin use started being captured in the UK and Swedish data sources (November 2016) and has and will be monitored annually thereafter until November 2020. The numbers were reported in annual interim reports in the 1st quarter of years 2017-2021 and the results of the interim reports were submitted to EMA by the Sponsor within the earliest corresponding PBRER. Initially, this study included two countries, the UK (CPRD GOLD) and Sweden, with follow-up until 31st December 2019. In order to increase the accumulated patient years and number of patients initiating the study drugs as well as accounting for the long latency period related to risk of malignancies, the study follow-up was first extended until 31st December, 2020 and Finnish national registers were included. Additionally, in this version of the protocol (Version 7.0) CPRD Aurum was included and the study period for both CPRD databases was extended to 31st December, 2021 in order to further increase the sample size and follow-up, and, consequently, study power.

<sup>2</sup> Observed IRs of 164.5, 104.1, and 58.0 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected number of empagliflozin initiators of 32,334, and matching ratio of 1:1.

<sup>3</sup> Observed IRs of 161.5, 86.8, and 71.6 per 100,000 person-years for UTC, bladder cancer, and renal cancer respectively, expected number of empagliflozin initiators of 18,269, and matching ratio of 1:2.

UK CPRD=The United Kingdom Clinical Practice Research Datalink

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8.6 DATA MANAGEMENT

Full audit trail starting from raw data obtained from register holders and ending with statistical tables and graphs in reports will be maintained. Data management, tabulations, graphics, and statistical modelling will be carried out with R data analyses language (http://www.r-project.org). R language is described more detailed in report "R: Regulatory Compliance and Validation Issues: A Guidance Document for the Use of R in Regulated Clinical Trial Environments" (http://www.r-project.org/doc/R-FDA.pdf). Source code of data management and data analyses is kept for inspection for five years after publication of results. The study may be inspected by the sponsor's study independent representative(s) or inspected by the competent authorities. A SEAP detailing all statistical analyses will be drawn and used as a basis for analysis.

Data from multiple country sources will be sent utilizing password protected media. All study related datasets will be stored in secured server environment. Access to data will be permitted only to study statisticians and data managers in line with the data permits. All data used for this study will be anonymous such that no study individual can be directly identified. Data will be regularly backed-up and stored in a separate secure location. All data and back-ups will be maintained within the EU.

### 8.7 DATA ANALYSIS

The final approach to data analysis will be presented in a separate SEAP to be developed prior to the start of data analysis. The SEAP will include a detailed algorithm for identifying T2D patients, detailed methods for covariate selection, checking for empirical equipoise, model checking for outcome models, methods for time-dependent exposure and time-varying confounding, the approaches for handling missing data, the assessment of the potential impact of unmeasured confounding, and the critical sensitivity analyses. The SEAP will be made available upon request to EMA and will be included or appended in the study report.

### 8.7.1 Main analysis

For the primary, secondary and further objectives, the main data analysis will be conducted in two stages: (i) construction of the PS-matched cohort by modelling the exposure to empagliflozin vs. DPP-4 inhibitors and (ii) estimating the effect of exposure to empagliflozin on the urinary tract (bladder, renal and other) cancers using aHRs and IRs compared to those exposed to DPP-4 inhibitors. Additional sensitivity analyses will be performed to validate the robustness of alternative definitions of outcome, exposure, covariates and reduction of bias due to matching.

### 8.7.1.1 Matching at index date

For all individuals, PS for the comparison of empagliflozin vs DPP-4 inhibitors will be computed at the index date as the probability to receive empagliflozin conditional on treatment and clinical history up to index date within each stratum. The PS will be estimated

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

using a binary logistic regression model. Depending on sample size, combination exposures with metformin will be accounted for through separate PS, stratification, or adjustment.

The selection of variables to be included in the PS models (see Section 8.3.3) will be based on scientific basis from previous studies, clinical/epidemiological significance and examination of exposure group differences in the distribution of each covariate. The covariates included in the PS model should ideally be associated with the outcomes of interest. Simulation studies show that variables that are unrelated to the exposure but are related to the outcome should always be included in the estimation of PS [R12-1913]. Inclusion of these variables increases the precision of the estimated effect of exposure without increasing bias. In contrast, inclusion of variables that are related to the exposure but not to the outcome can decrease precision of the estimated effect of exposure without decreasing bias. The variables listed in Annex 6 are potential candidates for inclusion in the PS model. Depending on sample size, combination exposures with metformin and treatment complexity (monotherapy, dual combination therapy, triple combination therapy) will be accounted for through separate PS, stratification, or adjustment.

Matching will be performed for empagliflozin initiators with patients initiating DPP-4 inhibitors within each country database. Matching will be carried out in several rounds to achieve the highest possible matching ratio given the available data in each country (up to 1:3 matching) [P12-07757]. In the first round of matching, for each empagliflozin initiating individual i with a particular index date TiE, all individuals initiating other DPP-4 inhibitors within three months before or after TiE will be chosen. Of these, one individual with the closest PS to that of i within a predefined PS interval will be selected as a match (Greedy matching method). The predefined PS interval will be calculated based on the standard deviation of the logit of PS ( $\delta$ ) multiplied by some coefficient k (say, k $\delta$ , when k=0.2). The value of the coefficient k will be calibrated to ensure at least 99% of those exposed to empagliflozin have matches from each comparator. The selected comparators are then removed from the pool of the possible comparators for further selection (sampling without replacement). Once the first round of matching is done, additional rounds of matching will be carried out to identify a second and possibly a third match for each already matched for each empagliflozin initiating individual (variable ratio matching with 1:3 as the maximum ratio). The number of matched DPP-4 inhibitors, and hence the overall matching ratio, will therefore be maximized within each country. Matching by time period, based on index dates, enables better control of time-varying confounders including changing prescription patterns for empagliflozin and potential confounding.

### 8.7.1.2 As-treated (AT) analysis

For the incident users of empagliflozin along with their respective matches, the primary analysis will be performed using the AT approach. This corresponds to censoring individuals who discontinue use of the index drug, i.e., either switch from the index drug to other drugs (empagliflozin, DPP-4 inhibitors, or other SGLT-2 inhibitors) during follow-up, or stop using the index drug (see Section 8.3.4).

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8.7.1.3 Population summary and descriptive analyses

Univariate and bivariate distribution of exposures, outcomes and relevant covariates will be presented using absolute and relative frequencies for categorical variables and summary measures for continuous variables (mean, standard deviation, median, min, max). Bivariate distributions for outcomes and covariates will be with reference to primary exposure definitions.

Absolute risks (IRs) for the defined outcomes will be estimated within each exposure category and key covariates using Poisson regression. The IRs will be presented along with 95% CIs. Other descriptive summaries such as number of events and person-time for calculating the IR will be included.

Kaplan-Meier plots, with 95% CIs, for survival probabilities will be presented for all urinary tract cancers, bladder cancers and renal cancers with primary exposures using the AT definition of follow-up times.

### 8.7.1.4 Comparative analyses

Relative risks (HRs) for the defined outcomes will be estimated using Cox models with time-varying covariates if model pre-requisites are fulfilled. HRs will be presented along with 95% CIs.

The Cox models will include the exposure and the comparator group within the model. This will account for multiple testing and for retaining same variables in variable selection (see Section 8.7.1.6). The models are defined in terms of covariates adjusted for in addition to the primary exposure: (i) baseline model with covariates adjusted for with values at index date (ii) model with time-dependent covariates wherein change in covariates over the follow-up period after index date are also incorporated into the model.

### **Country-specific analysis:**

The country-specific Cox models will be fit with single-country level datasets. The analyses will use datasets from the UK, Sweden, and Finland, separately.

### **Meta-analysis:**

Country-level effect sizes will be pooled using meta-analysis models to compute pooled effect size estimates. Prior to conducting meta-analyses, heterogeneity across the countries in terms of study design and conduct will be assessed. Specifically, the variability in population characteristics (including data availability), propensity score matching variables as well as propensity score balance will be examined.

Meta-analyses will be carried out for analyses where the country-level effect size is available for all three study countries. Pooled effect sizes will be estimated using random-effects models. The inverse-variance method will be used where appropriate.

# Protocol for non-interventional studies based on existing data BI Study Number 1245.97

c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Statistical heterogeneity between country-level estimates will be assessed using:

- Cochran's Q test
- I<sup>2</sup> statistic and its 95% CI
- The  $\tau^2$  statistic and its 95% CI

For each meta-analysis model, results will be presented in a forest plot including at least the following data:

- Data source.
- Effect size and 95% CI for each study included in the analysis (on a log scale).
- The weights allocated to each study.
- The combined estimated effect size with 95% CI (on a log scale) for the random-effects model.
- Value of Cochran's Q statistic, with the number of degrees of freedom and p-value.
- The proportion of variability explained by heterogeneity (I<sup>2</sup>).
- The between-study variance  $\tau^2$ .

If high levels of heterogeneity exist, the population characteristics and statistical models in the different country-level analyses will be reviewed and the possible source of heterogeneity discussed. A sensitivity analysis for the main analysis of the primary outcomes will be carried out using fixed-effect models to ascertain the effect of between-study heterogeneity on the meta-analysis result.

Further details regarding the meta-analysis models and heterogeneity will be defined in the study SEAP.

### 8.7.1.5 Variable selection

All potential confounders, exact and PS matching variables will enter the outcome model only after being selected using predefined variable selection criteria to be detailed in the SEAP.

### 8.7.1.6 Monitoring of accrual of empagliflozin users

Accrual of empagliflozin users, free or fixed-dose combinations with metformin, has been monitored starting at 24 months after use of empagliflozin was first captured in the UK and Swedish data sources (November 2016), and the numbers will be monitored annually until 2020. The purpose of this monitoring is to estimate the event rates for the outcomes of interest to confirm the event rates described in the literature and used in the sample size analyses. Finland was added in protocol version 5.0 and the final report will include data from the UK CPRD GOLD, CPRD Aurum, and National registers in Sweden and Finland.

The available power to estimate the association between empagliflozin use and the outcomes will be examined. If there is insufficient power (<80%) because, given the current event rates, the number of new users of empagliflozin accrued up to that point is too low to yield acceptable precision, decisions will be made about extending the length of the study period, the need to use additional country data sources, and/or changing the primary study design to a nested case-control study.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8.7.1.7 Handling of missing data

A high frequency of missing values is not expected for most variables, with the possible exception of lifestyle and laboratory parameters. For the medical history conditions/ comorbidities to be collected for inclusion in the PS, the absence of a code for a condition will be interpreted as an absence of the event. If a study variable is totally missing from a database (CPRD GOLD or Aurum, Sweden or Finland), it is excluded from the analysis of the pooled data. If a variable is missing for only some of the patients a missing data category will be added and utilized in the analysis.



Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



### 8.8 QUALITY CONTROL

The study will be conducted as specified in this protocol and SEAP. All revisions to the protocol shall be properly documented as protocol changes/amendments and when necessary, such protocol amendments will be delivered to register holder(s) whenever amendment(s) to the data permissions are required.

The study protocol has been written by following the Code of Conduct by the European Network of Centres for Pharmacoepidemiology and Pharmacovigilance (ENCePP) [R15-4870] that provides a set of rules and principles for post-authorisation studies with regard to the best practices and transparency, thereby promoting scientific independence of such studies. ENCePP is a project led by the EMA to further strengthen the post-authorisation monitoring of medicinal products in Europe by facilitating the conduct of multi-centre, independent, post-authorisation studies focusing on safety and on benefit/risk. The study will

# Protocol for non-interventional studies based on existing data BI Study Number 1245.97

c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

be registered to the ENCePP's E-register. The results of this study will also be published on the same site.

The study protocol also follows the key elements of the Guideline for Good Pharmacoepidemiology Practices by International Society for Pharmacoepidemiology [R11-4318], and the recent draft Guidance for Industry and FDA Staff "Best Practices for Conducting and Reporting Pharmacoepidemiologic Safety Studies Using Electronic Healthcare Data Sets" [R15-4859].

All programs for data management and data analyses will be written by study statistician(s). Ouality control check of these programs will be carried out by a statistician other than the one who writes the program. All processes from data management leading to dissemination of study results will undergo quality control checks for programs, result tables and written text. A detailed audit trail of all documents (programs, result tables, reports) along with quality control processes will be maintained.

#### LIMITATIONS OF THE RESEARCH METHODS 8.9

There are several methodological challenges to conducting epidemiological studies evaluating the comparative safety of glucose lowering medications [P12-13528, P14-17457, R14-4378, R13-1120, R10-6638].

The last (fifth) interim report (ANNEX 1) presented sample sizes of the study populations. It was noted that SGLT-2 inhibitor users were few and so that group was removed from analyses as stated in the amendments and updates, Section 4.

The actual use of prescribed or purchased drugs, especially oral glucose lowering medications cannot be verified with certainty. Drug exposure will be defined by algorithmic approaches based on the amount dispensed/prescribed in a prescription. This may be subject to misclassification. Sensitivity analyses will be performed to assess the impact of the exposure definitions on the main results.

The time-dependent nature of the exposure also creates a challenge due to time-dependent confounding. Although PS matching is used to control for imbalances between exposed and unexposed cohorts at the time of index date, other factors potentially associated with both exposure and outcome after index date are not controlled by PS matching. This may be tackled by use of causal models (e.g., marginal structural models, inverse-probability of weighting approach) as sensitivity analysis.

The AT approach used as the primary analysis may result in exclusion of cancer cases due to censoring at treatment discontinuation of the index drug. This will be addressed in sensitivity analyses as an ITT approach will be conducted. The ITT approach is conservative and is subject to exposure misclassification, but it ensures the evaluation of all cases occurring during the study period. For this reason, we will conduct sensitivity analyses considering a longer time period after treatment discontinuation. Finally, we will apply a 6-month lag

# Protocol for non-interventional studies based on existing data BI Study Number 1245.97

c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

period after the index date to the follow-up time in both the AT and ITT analyses to exclude subjects with only a short exposure time.

Determining the appropriate induction/promotion time window is challenging and typically only empirically based. Sensitivity analyses will evaluate a longer latency time window (12 months).

Although many variables may be included in the study, there will be relatively limited information (including age, sex, previous hospitalizations, chronic diseases) about risk factors connected to malignancies of UT from the available databases. For example, information on exposure to toxic chemicals is not available in the study databases. We attempt to control for the confounding bias by using baseline and time-dependent variables of potential confounders in the statistical analyses.

A potential limitation of using PS matching is that any exposed patient without a matched control would be excluded from the analyses. This will be tackled by applying a wider matching caliber for the PS for all unmatched cases after the first round of matching.

### 8.9.1 Bias

Potential source of difference in cancer incidence may arise due to channelling bias, detection bias and confounding. The channelling bias is addressed through both two-stage modelling approach wherein individuals are first matched on PS conditional on variables that affect exposure and outcome. Confounding will be minimized through model adjustment after carefully selecting variables using the variable selection criteria. However, there may be confounding due to unobserved variables and/or incomplete adjustment. Detection bias is inherent in cancer studies, especially those where the outcome is based on cancer notification. Although the notification is complete, early stages may go undetected. In studies including exposures with publicized safety concerns, diagnostic bias is also a concern, as patients with the exposure may be more likely to receive screenings for the outcome. The potential for diagnostic bias will be evaluated and addressed through consideration of the frequency of urine dipstick testing (as captured through albuminuria tests) and stage of cancer at the time of diagnosis (as more early-stage cancers in one group would be suggestive of diagnostic bias).

Bias due to definitions of exposure, definition of follow-up times and other relevant covariates will be addressed through sensitivity analyses. As mentioned in <u>Section 8.9</u>, the AT approach used as the primary analysis is subject to omission of cancer cases due do censoring after treatment switch or treatment discontinuation. An ITT approach will therefore be used in sensitivity analyses.

### 8.9.2 Generalizability

In the current study three population-based data sources (CPRD GOLD, CPRD Aurum, and Swedish and Finnish national registries) will be used. CPRD GOLD provides data entered by primary care practitioners in a routine clinical care setting and covers approximately 8.8% of

### Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1245.97

 c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

the UK population and CPRD Aurum about 13% of England population The patients are broadly representative of the UK population in terms of age, sex and ethnicity. In Sweden, the national registries cover practically all patients with T2D. In Finland, the coverage of the EMR data is approximately 26.7%, and study population is broadly generalizable. Therefore, the study results can be generalized to similar patients with T2D in other geographic settings, including most industrialized countries.
Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 9. PROTECTION OF HUMAN SUBJECTS

To ensure the full data protection of patients, all the research data in each country is anonymised. The implications of the General Data Protection Regulation (EU) 2016/679 on the national legislations, during the course of the study, will be considered. Approval from relevant Ethical/Research Review Boards will be required before conducting the study.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 10. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

Based on current guidelines from the International Society for Pharmacoepidemiology [R11-4318] and the EMA [R13-1970], non-interventional studies such as the one described in this protocol, conducted using medical chart reviews or electronic claims and health care records, do not require expedited reporting of suspected adverse events/reactions. Specifically, as stated in section VI.C.1.2.1 of Guideline on Good Pharmacovigilance Practices (GVP), Module VI – Management and Reporting of Adverse Reactions to Medicinal Products, for non-interventional study designs, which are based on use of secondary data, reporting of adverse reactions is not required.

The data generated in the course of the study will be monitored by the BI responsible person.

When an observation is identified that may qualify as a special safety issue or that may have implications for the benefit-risk balance of empagliflozin, appropriate BI functions will be notified according to BI standard operating procedures.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 11. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

Study reports will be prepared using a template following the Guideline on Good Pharmacovigilance Practices (GVP), Module VIII, Section B.6.3 [R13-5420]. The principal and co-investigators will write the annual interim reports and the final study report. The reports will be delivered to the Sponsor. The Sponsor will submit the interim and the final reports to EMA in line with the milestones (see Section 5) and report the results within the earliest corresponding PSURs; the final report will be submitted to the EMA as a type II variation. The study results will be published in the EU PASS registry.

The principal and co-investigators will co-author scientific manuscript(s) of the results to be published. The publication strategy is defined in the research agreement between the principal investigators and the Sponsor. A summary of the main results of the study, whether positive or negative and including results from prematurely terminated studies, will always be made available to the public. Per Section V of Guidelines for Good Pharmacoepidemiology Practices (GPP) [R11-4318] and the Guideline on Good Pharmacovigilance Practices, Module VIII, Section B.7 [R13-5420]. The outcome of a study will always be presented in an objective and truthful manner providing a comprehensive and accurate description of the findings. In no way shall the interpretation and presentation of the results be aimed towards any commercial, financial or personal interests.

The Sponsor is entitled to view the final results and interpretations thereof prior to submission for publication and to comment in advance of submission as agreed in the research contract and without unjustifiably delaying the publication.

### 12. REFERENCES

#### 12.1 PUBLISHED REFERENCES

P12-07757 Rassen JA, Shelat AA, Myers J, Glynn RJ, Rothman KJ, Schneeweiss S. Oneto-many propensity score matching in cohort studies. Pharmacoepidemiol Drug Saf 2012; 21(Suppl 2); 69-80. Lo Re V, 3rd, Haynes K, Ming EE, Wood Ives J, Horne LN, Fortier K, et al. P12-13528 Safety of saxagliptin: rationale for and design of a series of postmarketing observational studies. Pharmacoepidemiol Drug Saf 2012; 21 (11): 1202-15. P14-16383 Macedo AF, Douglas I, Smeeth L, Forbes H, Ebrahim S. Statins and the risk of type 2 diabetes mellitus: cohort study using the UK clinical practice pesearch datalink. BMC Cardiovasc Disord. 2014; 14: 85. NICE. Type 2 diabetes: the management of type 2 diabetes. NICE clinical P14-17374 guideline 87. National Institute for Health and Care Excellence; 2014. Available at: website: nice.org.uk/guidance/cg87/resources/guidance-type-2diabetes-pdf. Accessed 09 October 2014. Rawson NS. Review of the quality of observational studies of the association P14-17457 between rosiglitazone and acute myocardial infarction. J Popul Ther Clin Pharmacol 2014; 21 (2): e214-32. Tuomi T, Antikainen A, Hokasalo M, Härmä-RodriguezS, Ilanne-Parikka P et P19-01624 al., Finnish Medical Society Duodecim. Diabetes. Current Care Guideline, 2018. Statistical database Kelasto [Internet]. The Social Insurance Institution of P19-01956 Finland [cited 2019 August 21]. Available from: http://raportit.kela.fi/ibi\_apps/WFServlet?IBIF\_ex=NIT137AL&YKIELI=E Boehringer Ingelheim. Endocrinologic and metabolic drugs advisory P19-01957 committee briefing document. EMPA-REG OUTCOME® Trial. 19 May 2016. The CANVAS Program (CANagliflozin cardioVascular Assessment Study). P19-07186 Conference presentation at American Diabetes Association (ADA) 77th Scientific Sessions. Available from: https://www.georgeinstitute.org/sites/default/files/canvas-study-results-ada-2017.pdf R10-6494 Vigneri P, Frasca F, Sciacca L, Pandini G, Vigneri R. Diabetes and cancer. Endocrine-Related Cancer, 2009; 16: 1103-23. Lindbald P, Chow WH, Chan J, Bergström A, Wolk A, et al. The role of R10-6630 diabetes mellitus in the aetiology of renal cell cancer. Diabetologia 1999; 42: 107-12. Giovannucci E, Harlan DM, Archer MC, Bergenstal RM, Gapstur SM, Habel R10-6638 LA, Pollak M, Regensteiner JG, Yee D. Diabetes and cancer: a consensus report. Diabetes Care 2010; 33 (7): 1674-1685. ISPE, International Society for Pharmacoepidemiology. Guidelines for Good R11-4318

Pharmacoepidemiological Practices. Revision 2: April 2007. www.pharmacoepi.org/resources/guidelines 08027.cfm.

| R11-5320 | Gonzalez EL, Johansson S, Wallander MA, Rodriguez LA. Trends in the prevalence and incidence of diabetes in the UK: 1996-2005. J Epidemiol |
|---|---|
| R12-0368 | Community Health 2009; 63 (4): 332-6.<br>Larsson SC, Andersson SO, Johansson JE, Wolk A. Diabetes mellitus, body size and bladder cancer risk in a prospective study of Swedish men. Eur J |
| | Cancer 44:2655-2660. |
| R12-0469 | Larsson SC, Orsini N, Brismar K, Wolk A. Diabetes mellitus and risk of bladder cancer: a meta-analysis. Diabetologia 2006; 49: 2819-23. |
| R12-1334 | Carstensen B, Witte DR, Friis S. Cancer occurrence in Danish diabetic patients: duration and insulin effects. Diabetologia 2012; 55:948-958. |
| R12-1620 | EMA. European Medicines Agency recommends suspension of Avandia, Avandamet and Avaglim (press release). 23 September 2010. Available at: website: ema.europa.eu/ema/index.jsp?curl = |
| | pages/news_and_events/news/2010/09/news_detail_001119.jsp∣ = WC0b01ac058004d5c1. Accessed 09 October 2014. |
| R12-1913 | Brookhart MA, Schneeweiss S, Rothman KJ, Glynn RJ, Avorn J, Sturmer T. Variable selection for propensity score models. Am J Epidemiol. 2006 Jun 15; 163 (12): 1149-56. |
| R12-2439 | Onitilo AA, Engel JM, Glurich I, Stankowski RV, Williams GM, Doi SA Diabetes and cancer I: risk, survival, and implications for screening. Cancer |
| R13-1120 | Causes Control 2012; 23:967-981. Schneeweiss S. A basic study design for expedited safety signal evaluation based on electronic healthcare data. Pharmacoepidemiol Drug Saf 2010; 19 |
| R13-1812 | (8): 858-68. Bao C, Yang X, Xu W, Luo H, Xu Z, Su C, Qi X. Diabetes mellitus and incidence and mortality of kidney cancer: a meta-analysis. J Diabetes |
| R13-1970 | Complications 2013;27:357–364. EMA. Guideline on good pharmacovigilance practices (GVP). Module VI – Management and reporting of adverse reactions to medicinal products. European Medicines Agency; 22 June 2012. Available at: website: |
| R13-5134 | emea.europa.eu/docs/en_GB/document_library/Scientific_guideline/2012/06/WC500129135.pdf. Accessed 7 February 2013. NICE. Dapagliflozin in combination therapy for treating type 2 diabetes. NICE technology appraisal guidance 288. National Institute for Health and Care |
| R13-5420 | Excellence; 2013. Available at: website: nice.org.uk/guidance/ta288/resources/guidance-dapagliflozin-in-combination-therapy-for-treating-type2-diabetes-pdf. Accessed 09 October 2014. EMA. Guideline on good pharmacovigilance practices (GVP). Module VIII – Post-authorisation safety studies. European Medicines Agency; 9 July 2012. |
| | Available at website |

emea.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2012/06/

WC500129137.pdf. Accessed 7 February 2013.

- R14-4378 Patorno E, Patrick AR, Garry EM, Schneeweiss S, Gillet VG, Bartels DB, et al. Observational studies of the association between glucose-lowering medications and cardiovascular outcomes: addressing methodological limitations. Diabetologia 2014; 57 (11): 2237-50.
- R14-4617 Boehringer Ingelheim International GmbH. Jardiance (empagliflozin) summary of product characteristics. 2014. Available at: website: ema.europa.eu/ema/index.jsp?curl = pages/medicines/human/medicines/002677/human\_med\_001764.jsp&mid = WC0b01ac058001d124. Accessed 09 October 2014.
- R14-5244 Leal I, Romio SA, Schuemie M, Oteri A, Sturkenboom M, Trifiro G. Prescribing pattern of glucose lowering drugs in the United Kingdom in the last decade: a focus on the effects of safety warnings about rosiglitazone. Br J Clin Pharmacol 2013; 75 (3): 861-8.
- Morgan CL, Poole CD, Evans M, Barnett AH, Jenkins-Jones S, Currie CJ. What next after metformin? A retrospective evaluation of the outcome of second-line, glucose-lowering therapies in people with type 2 diabetes. J Clin Endocrinol Metab 2012; 97 (12): 4605-12.
- R15-4856 Kreiger N, Marrett LD, Dodds L, Hilditch S, Darlington GA. Risk factors for renal cell carcinoma: results of a population-based case-control study. Cancer Causes Control 1993; 4(2):101-110.
- R15-4857 Korhonen P, Malila N, Pukkala E, Teppo L, Albanes D, Virtamo J. The Finnish Cancer Registry as Follow-Up Source of a Large Trial Cohort. Acta Oncologica. 2002; 41: 381-388.
- R15-4858 Jansson SPO, Fall K, Brus O, Magnuson A, Wändell P, Östgren CJ, Rolandsson O. Prevalence and incidence of diabetes mellitus: a nationwide population-based pharmaco-epidemiological study in Sweden. Diab Med 2015.
- R15-4859 FDA, Food and Drug Administration. Guidance for Industry and FDA Staff. Best Practices for Conducting and Reporting Pharmacoepidemiologic Safety Studies Using Electronic Healthcare Data Sets. February 2011. www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM243537.pdf
- Forman D, Bray F, Brewster DH et al., eds [Internet]. Cancer Incidence in Five Continents, Vol. X (electronic version) Lyon, IARC [cited 2015 June 23]. Available from: http://ci5.iarc.fr/Default.aspx
- Furu K, Wettermark B, Andersen M et al. The Nordic countries as a cohort for pharmacoepidemiological research. Basic Clin. Pharmacol. Toxicol. 2010, 106:86-94.
- R15-4862 Dregan A, Moller H, Murray-Thomas T and Gulliford MC. Validity of cancer diagnosis in a primary care database compared with linked cancer registrations in England. Population-based cohort study. Cancer Epidemiol. Elsevier Ltd; 2012 Oct;36(5):425–9.
- R15-4863 Chow WH, Lindblad P, Gridley G, Nyren O, McLaughlin JK, Linet MS, Pennello GA, Adami HO, Fraumeni JF. Risk of urinary tract cancers following kidney or ureter stones. J Natl Cancer Inst 1997; 89(19):1453-1457.

| R15-4864 | Boggon R, van Staa TP, Chapman M, Gallagher AM, Hammad TA, Richards MA. Cancer recording and mortality in the General Practice Research Database and linked cancer registries. Pharmacoepidemiol Drug Saf. 2013 Feb; 22(2): 168–75. |
|---|---|
| R15-4865 | Boffetta P, Jourenkova N, Gustavsson P. Cancer risk from occupational and environmental exposure to polycyclic aromatic hydrocarbons. Cancer Causes Control 1997; 8(3):444-472. |
| R15-4866 | Burger M, Catto JWF, Dalbagni G, Grossman HB, Herr H, Karakiewicz P, Kassouf W, Kiemeney LA, Vecchia C la, Shariat S, Lotan Y. Epidemiology and risk factors of urothelial bladder cancer. Eur Urol 2013; 63(2):234-241. |
| R15-4867 | Barlow L, Westergren K, Holmberg L and Talbäck M. The completeness of the Swedish Cancer Register – a sample survey for year 1998. Acta Oncologica. 2009; 48: 27-33. |
| R15-4868 | Zeegers MPA, Tan FE, Dorant E, Brandt PA van den. The impact of characteristics of cigarette smoking on urinary tract cancer risk: a meta-analysis of epidemiologic studies. Cancer 2000; 89(3):630-639. |
| R15-4869 | Wideroff L, Gridley G, Mellemkjaer L et al. Cancer incidence in a population-based cohort of patients hospitalized with diabetes mellitus in Denmark. J. Natl. Cancer Inst. 1997; 89: 1360-5. |
| R15-4870 | ENCePP. The ENCePP Code of Conduct for Scientific Independence and Transparency in the Conduct of Pharmacoepidemiological and Pharmacovigilance Studies. 21 November 2011, EMA/929209/2011. www.encepp.eu/code of conduct/documents/CodeofConduct Rev2.pdf |
| R15-4871 | Teppo L, Pukkala E and Lehtonen M. Data quality and quality control of a population-based cancer registry. Acta Oncologica. 1994; 33: 365-369. |
| R15-4873 | NORDCAN Register [Internet]. Association of the Nordic Cancer Registries [cited 2015 June 18]. Available from: http://www-dep.iarc.fr/NORDCAN/english/frame.asp |
| R16-1231 | Herrett et al. Data Resource Profile: Clinical Practice Research Datalink (CPRD). Int J Epidemiol. 2015 44:827-36. |
| R16-2539 | Murchie P, Campbell NC, Delaney EK, Dinant GJ, Hannaford PC et al. Comparing Diagnostic delay in Cancer: a cross-sectional study in three European Countries with primary care. led health care systems. Fam Pract. 2012 29: 69-78. |
| R17-0153 | Boehringer Ingelheim International GmbH. Synjardy (empagliflozin, metformin hydrochloride) Summary of Product Characteristics. Available at: https://www.ema.europa.eu/en/documents/product-information/synjardy-epar-product-information_en.pdf. Accessed 21 August 2019 |
| R19-1534 | Wolf et al. Data resource profile: Clinical Practice Research Datalink (CPRD) Aurum. Int J Epidemiol. 2019 Mar 11. pii: dyz034. |
| R19-2814 | Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med 2019;380:347–357. |

c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

R19-2928 CPRD linked data [Internet, page last reviewed 8 August 2019]. Clinical Practice Research Datalink [cited 2019 Aug 21]. Available from: https://www.cprd.com/linked-data

## 12.2 UNPUBLISHSED REFERENCES

Not Applicable

## 13. ANNEXURE

## ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

| Number | Document<br>number | Date | Title |
|---|---|---|---|
| 1 | c27031418-01 | 08 June 2021 | Post-authorisation safety study to assess the risk of urinary tract malignancies in relation to empagliflozin exposure in patients with type 2 diabetes: a multidatabase European study – Fifth monitoring interim report |

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS



Doc.Ref. EMA/540136/2009



#### **ENCePP Checklist for Study Protocols (Revision 4)**

Adopted by the ENCePP Steering Group on 15/10/2018

The European Network of Centres for Pharmacoepidemiology and Pharmacovigilance (ENCePP) welcomes innovative designs and new methods of research. This Checklist has been developed by ENCePP to stimulate consideration of important principles when designing and writing a pharmacoepidemiological or pharmacovigilance study protocol. The Checklist is intended to promote the quality of such studies, not their uniformity. The user is also referred to the ENCePP Guide on Methodological Standards in Pharmacoepidemiology, which reviews and gives direct electronic access to guidance for research in pharmacoepidemiology and pharmacovigilance.

For each question of the Checklist, the investigator should indicate whether or not it has been addressed in the study protocol. If the answer is "Yes", the section number of the protocol where this issue has been discussed should be specified. It is possible that some questions do not apply to a particular study (for example, in the case of an innovative study design). In this case, the answer 'N/A' (Not Applicable) can be checked, and the "Comments" field included for each section should be used to explain why. The "Comments" field can also be used to elaborate on a "No" answer.

This Checklist should be included as an Annex by marketing authorisation holders when submitting the protocol of a non-interventional post-authorisation safety study (PASS) to a regulatory authority (see the Guidance on the format and content of the protocol of non-interventional postauthorisation safety studies). The Checklist is a supporting document and does not replace the format of the protocol for PASS presented in the Guidance and Module VIII of the Good pharmacovigilance practices (GVP).

### Study title:

Post-authorisation safety study to assess the risk of urinary tract malignancies in relation to empagliflozin exposure in patients with type 2 diabetes: a multi-database European study

EU PAS Register® number: EUPAS16424 Study reference number (if applicable): c03856813-08

| Section 1: Milestones | | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| 1.1 | Does the protocol specify timelines for | | | | |
| | 1.1.1 Start of data collection <sup>1</sup> | $\boxtimes$ | | | 5 |
| | 1.1.2 End of data collection <sup>2</sup> | $\boxtimes$ | | | 5 |
| | 1.1.3 Progress report(s) | | | $\boxtimes$ | |

Date from which information on the first study is first recorded in the study dataset or, in the case of secondary use of data, the date from which

data extraction starts.

<sup>2</sup> Date from which the analytical dataset is completely available.

| Secti | on 1: Milestones | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| | 1.1.4 Interim report(s) | $\boxtimes$ | | | 5 |
| | 1.1.5 Registration in the EU PAS Register® | $\boxtimes$ | | | 5 |
| | 1.1.6 Final report of study results. | $\boxtimes$ | | | 5 |
| omn | nents: | | | | |
| Sect | on 2: Research question | Yes | No | N/A | Section<br>Number |
| 2.1 | Does the formulation of the research question and objectives clearly explain: | $\boxtimes$ | | | |
| | 2.1.1 Why the study is conducted? (e.g. to address an important<br>public health concern, a risk identified in the risk management plan, an<br>emerging safety issue) | $\boxtimes$ | | | 6 |
| | 2.1.2 The objective(s) of the study? | $\boxtimes$ | | | 7 |
| | 2.1.3 The target population? (i.e. population or subgroup to whom the study results are intended to be generalised) | $\boxtimes$ | | | 8.2.1 |
| | 2.1.4 Which hypothesis(-es) is (are) to be tested? | | | $\boxtimes$ | |
| | 2.1.5 If applicable, that there is no a priori hypothesis? | | | $\boxtimes$ | |
| | on 3: Study design | Yes | No | N/A | Section<br>Number |
| 3.1 | Is the study design described? (e.g. cohort, case-control, cross-<br>sectional, other design) | $\boxtimes$ | | | 8.1 |
| 3.2 | Does the protocol specify whether the study is based on primary, secondary or combined data collection? | $\boxtimes$ | | | 8.1 |
| 3.3 | Does the protocol specify measures of occurrence? (e.g., rate, risk, prevalence) | $\boxtimes$ | | | 8.1 |
| 3.4 | Does the protocol specify measure(s) of association? (e.g. risk, odds ratio, excess risk, rate ratio, hazard ratio, risk/rate difference, number needed to harm (NNH)) | $\boxtimes$ | | | 8.1 |
| 3.5 | Does the protocol describe the approach for the collection and reporting of adverse events/adverse reactions? (e.g. adverse events that will not be collected in case of primary data collection) | $\boxtimes$ | | | 10 |
| omn | nents: | | | | |
| Secti | on 4: Source and study populations | Yes | No | N/A | Section<br>Number |
| 4.1 | Is the source population described? | $\boxtimes$ | | | 8.2 |
| 4.2 | Is the planned study population defined in terms of: | | | | 8 |
| | 4.2.1 Study time period | $\boxtimes$ | | | 8.2.2 |
| | 4.2.2 Age and sex | $\boxtimes$ | | | 8.2.5 |
| | 4.2.2 Age and sex | 1 | | 1 - | 0.0.1 |
| | 4.2.3 Country of origin | $\boxtimes$ | | | 8.2.1 |
| | (and the original of the control of | $\boxtimes$ | | | 8.2.1 |

| Section 4: Source and study populations | | | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| 4.3 | Does the protocol define how the study population will be sampled from the source population? (e.g. event or inclusion/exclusion criteria) | | | | 8.2.5 |
| omm | ents: | | | | |
| Secti | on 5: Exposure definition and measurement | Yes | No | N/A | Section<br>Number |
| 5.1 | Does the protocol describe how the study exposure is defined<br>and measured? (e.g. operational details for defining and categorising<br>exposure, measurement of dose and duration of drug exposure) | $\boxtimes$ | | | 8.3.1 |
| 5.2 | Does the protocol address the validity of the exposure measurement? (e.g. precision, accuracy, use of validation sub-study) | $\boxtimes$ | | | 8.3.1 |
| 5.3 | Is exposure categorised according to time windows? | $\boxtimes$ | | | 8.3.1 |
| 5.4 | Is intensity of exposure addressed?<br>(e.g. dose, duration) | $\boxtimes$ | | | 8.3.1 |
| 5.5 | Is exposure categorised based on biological mechanism of action and taking into account the pharmacokinetics and pharmacodynamics of the drug? | | $\boxtimes$ | | |
| 5.6 | Is (are) (an) appropriate comparator(s) identified? | $\boxtimes$ | | | 8.3.1 |
| | on 6: Outcome definition and measurement | 13813119793 | SAMPLINGS | 100 CO | |
| | | | | | Number |
| 6.1 | Does the protocol specify the primary and secondary (if applicable) outcome(s) to be investigated? | $\boxtimes$ | | | Number<br>8.3.2 |
| 6.1 | | $\boxtimes$ | | | |
| 0.3% | applicable) outcome(s) to be investigated? Does the protocol describe how the outcomes are defined and | | | | 8.3.2 |
| 6.2 | applicable) outcome(s) to be investigated? Does the protocol describe how the outcomes are defined and measured? Does the protocol address the validity of outcome measurement? (e.g. precision, accuracy, sensitivity, specificity, positive | | | | 8.3.2<br>8.3.2 |
| 6.2 | applicable) outcome(s) to be investigated? Does the protocol describe how the outcomes are defined and measured? Does the protocol address the validity of outcome measurement? (e.g. precision, accuracy, sensitivity, specificity, positive predictive value, use of validation sub-study) Does the protocol describe specific outcomes relevant for Health Technology Assessment? (e.g. HRQoL, QALYS, DALYS, health care services utilisation, burden of disease or treatment, compliance, disease management) | | | | 8.3.2<br>8.3.2 |
| 6.2<br>6.3<br>6.4 | applicable) outcome(s) to be investigated? Does the protocol describe how the outcomes are defined and measured? Does the protocol address the validity of outcome measurement? (e.g. precision, accuracy, sensitivity, specificity, positive predictive value, use of validation sub-study) Does the protocol describe specific outcomes relevant for Health Technology Assessment? (e.g. HRQoL, QALYS, DALYS, health care services utilisation, burden of disease or treatment, compliance, disease management) ents: | | | | 8.3.2<br>8.3.2 |
| 6.2<br>6.3<br>6.4 | applicable) outcome(s) to be investigated? Does the protocol describe how the outcomes are defined and measured? Does the protocol address the validity of outcome measurement? (e.g. precision, accuracy, sensitivity, specificity, positive predictive value, use of validation sub-study) Does the protocol describe specific outcomes relevant for Health Technology Assessment? (e.g. HRQoL, QALYS, DALYS, health care services utilisation, burden of disease or treatment, compliance, disease management) | | | □ | 8.3.2<br>8.3.2 |
| 6.2<br>6.3<br>6.4 | applicable) outcome(s) to be investigated? Does the protocol describe how the outcomes are defined and measured? Does the protocol address the validity of outcome measurement? (e.g. precision, accuracy, sensitivity, specificity, positive predictive value, use of validation sub-study) Does the protocol describe specific outcomes relevant for Health Technology Assessment? (e.g. HRQoL, QALYS, DALYS, health care services utilisation, burden of disease or treatment, compliance, disease management) ents: | | | | 8.3.2<br>8.3.2<br>8.3.2 |
| 6.2<br>6.3<br>6.4<br>Comm | applicable) outcome(s) to be investigated? Does the protocol describe how the outcomes are defined and measured? Does the protocol address the validity of outcome measurement? (e.g. precision, accuracy, sensitivity, specificity, positive predictive value, use of validation sub-study) Does the protocol describe specific outcomes relevant for Health Technology Assessment? (e.g. HRQoL, QALYS, DALYS, health care services utilisation, burden of disease or treatment, compliance, disease management) ents: on 7: Bias Does the protocol address ways to measure confounding? (e.g. | Yes | □ □ □ No | N/A | 8.3.2<br>8.3.2<br>8.3.2<br>Section<br>Number |

| Section | on 8: Effect measure modification | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| 3.1 | Does the protocol address effect modifiers? (e.g. collection of data<br>on known effect modifiers, sub-group analyses, anticipated direction of effect) | $\boxtimes$ | | | 8.7.2 |
| mm | ents: | | | | |
| Section | on 9: Data sources | Yes | No | N/A | Section<br>Number |
| 0.1 | Does the protocol describe the data source(s) used in the study for the ascertainment of: | | | | |
| | 9.1.1 Exposure? (e.g. pharmacy dispensing, general practice prescribing, claims data, self-report, face-to-face interview) | $\boxtimes$ | | | 8.4 |
| | 9.1.2 Outcomes? (e.g. clinical records, laboratory markers or values, claims data, self-report, patient interview including scales and questionnaires, vital statistics) | $\boxtimes$ | | | 8.4 |
| | 9.1.3 Covariates and other characteristics? | $\boxtimes$ | | | 8.4 |
| 0.2 | Does the protocol describe the information available from the data source(s) on: | | 4 | | |
| | 9.2.1 Exposure? (e.g. date of dispensing, drug quantity, dose, number of days of supply prescription, daily dosage, prescriber) | $\boxtimes$ | | | 8.4 |
| | 9.2.2 Outcomes? (e.g. date of occurrence, multiple event, severity measures related to event) | | | | 8.4 |
| | <ol> <li>Covariates and other characteristics? (e.g. age, sex, clinical<br/>and drug use history, co-morbidity, co-medications, lifestyle)</li> </ol> | | | | 8.4 |
| 0.3 | Is a coding system described for: | | | | |
| | 9.3.1 Exposure? (e.g. WHO Drug Dictionary, Anatomical Therapeutic Chemical (ATC) Classification System) | $\boxtimes$ | | | 8.3 |
| | 9.3.2 Outcomes? (e.g. International Classification of Diseases (ICD),<br>Medical Dictionary for Regulatory Activities (MedDRA)) | $\boxtimes$ | | | 8.3 |
| | 9.3.3 Covariates and other characteristics? | $\boxtimes$ | | | 8.3 |
| 0.4 | Is a linkage method between data sources described? (e.g. based on a unique identifier or other) | $\boxtimes$ | | | 8.3 |
| mm | ents: | | | | |
| Section | on 10: Analysis plan | Yes | No | N/A | Section<br>Number |
| 0.1 | Are the statistical methods and the reason for their choice described? | $\boxtimes$ | | | 8.7 |
| 0.2 | Is study size and/or statistical precision estimated? | $\boxtimes$ | | | 8.7 |
| 0.3 | Are descriptive analyses included? | $\boxtimes$ | | | 8.7 |
| 0.4 | Are stratified analyses included? | $\boxtimes$ | | | 8.7 |
| 0.5 | Does the plan describe methods for analytic control of confounding? | $\boxtimes$ | | | 8.7 |
| 0.6 | Does the plan describe methods for analytic control of outcome misclassification? | $\boxtimes$ | | | 8.7 |
| 0.7 | Does the plan describe methods for handling missing data? | $\boxtimes$ | | | 8.7 |
| | Are relevant sensitivity analyses described? | $\boxtimes$ | | | 8.7 |

| Section | on 11: Data management and quality control | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| 11.1 | Does the protocol provide information on data storage?<br>(e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) | $\boxtimes$ | | | 8.6 |
| 11.2 | Are methods of quality assurance described? | $\boxtimes$ | | | 8.8 |
| 11.3 | Is there a system in place for independent review of study results? | | $\boxtimes$ | | |
| omm | ents: | * | | | |
| Section | on 12: Limitations | Yes | No | N/A | Section<br>Number |
| 12.1 | Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). | | | | 8.9<br>8.9<br>8.9 |
| 12.2 | Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) | $\boxtimes$ | | | 8.4 |
| Comme | ents: | | | | |
| Section | on 13: Ethical/data protection issues | Yes | No | N/A | Section<br>Number |
| 13.1 | Have requirements of Ethics Committee/ Institutional Review Board been described? | | | | 9 |
| 13.2 | Has any outcome of an ethical review procedure been addressed? | | $\boxtimes$ | | |
| 13.3 | Have data protection requirements been described? | $\boxtimes$ | | | 9 |
| Comme | ents: | | | | |
| Section | on 14: Amendments and deviations | Yes | No | N/A | Section<br>Number |
| 14.1 | Does the protocol include a section to document amendments and deviations? | $\boxtimes$ | | | 4 |
| Commo | ents: | | XV. | *** | |
| Section | on 15: Plans for communication of study results | Yes | No | N/A | Section |
| 15.1 | Are plans described for communicating study results (e.g. to regulatory authorities)? | $\boxtimes$ | | | Number<br>11 |
| | regulatory authorities): | | | | |

| Section 15: Plans for communication of study results | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|
| 15.2 Are plans described for disseminating study results externally, including publication? | $\boxtimes$ | | | 11 |
| Comments: | | | | |
| we s s wa s | | | | |
| Name of the main author of the protocol: | | | | |
| Name of the main author of the protocol: Date: 27/January/2022 | | | | |
| • | | | | |

## ANNEX 3. READ CODES TO IDENTIFY TYPE 2 DIABETES

The codes will be updated for the data application.

| Read code | Description |
|-----------|-------------------------------------------------------------|
| 9OL00 | Diabetes monitoring admin |
| 66A00 | Diabetic monitoring |
| 66AS.00 | Diabetic annual review |
| C1000 | Diabetes mellitus |
| 9N1Q.00 | Seen in diabetic clinic |
| C10F.00 | Type 2 diabetes mellitus |
| 9OL4.00 | Diabetes monitoring 1st letter |
| 66A2.00 | Follow-up diabetic assessment |
| 9NND.00 | Under care of diabetic foot screener |
| 66AP.00 | Diabetes: practice programme |
| 9OL1.00 | Attends diabetes monitoring |
| 66A4.00 | Diabetic on oral treatment |
| 68A7.00 | Diabetic retinopathy screening |
| 66AZ.00 | Diabetic monitoring NOS |
| 66AJ.00 | Diabetic - poor control |
| C100112 | Non-insulin dependent diabetes mellitus |
| 66Ac.00 | Diabetic peripheral neuropathy screening |
| 9OL5.00 | Diabetes monitoring 2nd letter |
| 66A3.00 | Diabetic on diet only |
| 66Aq.00 | Diabetic foot screen |
| C109.00 | Non-insulin dependent diabetes mellitus |
| F420.00 | Diabetic retinopathy |
| 13B1.00 | Diabetic diet |
| 9OLA.00 | Diabetes monitor. check done |
| 7L19800 | Subcutaneous injection of insulin |
| 66AR.00 | Diabetes management plan given |
| 9h42.00 | Excepted from diabetes quality indicators: Informed dissent |
| 2G5E.00 | O/E - Right diabetic foot at low risk |
| 66A5.00 | Diabetic on insulin |

| Read code | Description |
|-----------|------------------------------------------------------------|
| 2G5I.00 | O/E - Left diabetic foot at low risk |
| 9h41.00 | Excepted from diabetes qual indicators: Patient unsuitable |
| F420000 | Background diabetic retinopathy |
| 9N4I.00 | DNA - Did not attend diabetic clinic |
| 66AI.00 | Diabetic - good control |
| C109.12 | Type 2 diabetes mellitus |
| 66AQ.00 | Diabetes: shared care programme |
| 66AD.00 | Fundoscopy - diabetic check |
| 8BL2.00 | Patient on maximal tolerated therapy for diabetes |
| 1434.00 | H/O: diabetes mellitus |
| 9OL6.00 | Diabetes monitoring 3rd letter |
| 66Ai.00 | Diabetic 6 month review |
| 9N1v.00 | Seen in diabetic eye clinic |
| 8CA4100 | Pt advised re diabetic diet |
| 2BBP.00 | O/E - right eye background diabetic retinopathy |
| 2BBQ.00 | O/E - left eye background diabetic retinopathy |
| 8B31.00 | Diabetes medication review |
| 66A9.00 | Understands diet - diabetes |
| 66Ab.00 | Diabetic foot examination |
| 42W00 | Hb. A1C - diabetic control |
| 66AU.00 | Diabetes care by hospital only |
| 9NM0.00 | Attending diabetes clinic |
| 8H7r.00 | Refer to diabetic foot screener |
| 8I3X.00 | Diabetic retinopathy screening refused |
| 2G5F.00 | O/E - Right diabetic foot at moderate risk |
| 2G5J.00 | O/E - Left diabetic foot at moderate risk |
| 66A1.00 | Initial diabetic assessment |
| F420400 | Diabetic maculopathy |
| 66AW.00 | Diabetic foot risk assessment |
| 90LA.11 | Diabetes monitored |
| 13AB.00 | Diabetic lipid lowering diet |

| Read code | Description |
|-----------|-------------------------------------------------------------|
| 2BBM.00 | O/E - diabetic maculopathy absent both eyes |
| ZC2C800 | Dietary advice for diabetes mellitus |
| C100100 | Diabetes mellitus, adult onset, no mention of complication |
| 66Ao.00 | Diabetes type 2 review |
| 9OL8.00 | Diabetes monitor.phone invite |
| 9N4p.00 | Did not attend diabetic retinopathy clinic |
| 9N1i.00 | Seen in diabetic foot clinic |
| 14P3.00 | H/O: insulin therapy |
| C101.00 | Diabetes mellitus with ketoacidosis |
| 66A8.00 | Has seen dietician - diabetes |
| 66AT.00 | Annual diabetic blood test |
| C10FJ00 | Insulin treated Type 2 diabetes mellitus |
| 9OL3.00 | Diabetes monitoring default |
| 66AV.00 | Diabetic on insulin and oral treatment |
| 66A7.00 | Frequency of hypo. attacks |
| 9OL11 | Diabetes clinic administration |
| 66AA.11 | Injection sites - diabetic |
| 66AH000 | Conversion to insulin |
| 8CS0.00 | Diabetes care plan agreed |
| 2G5G.00 | O/E - Right diabetic foot at high risk |
| 66AH.00 | Diabetic treatment changed |
| 2G5K.00 | O/E - Left diabetic foot at high risk |
| 9OLD.00 | Diabetic patient unsuitable for digital retinal photography |
| F372.12 | Diabetic neuropathy |
| F420600 | Non-proliferative diabetic retinopathy |
| C106.12 | Diabetes mellitus with neuropathy |
| 9OL7.00 | Diabetes monitor. verbal invite |
| C106.00 | Diabetes mellitus with neurological manifestation |
| 8H4F.00 | Referral to diabetologist |
| 8I3W.00 | Diabetic foot examination declined |
| 68A9.00 | Diabetic retinopathy screening offered |

| Read code | Description |
|-----------|-------------------------------------------------------------|
| 13AC.00 | Diabetic weight reducing diet |
| F420100 | Proliferative diabetic retinopathy |
| 66AY.00 | Diabetic diet - good compliance |
| C10FM00 | Type 2 diabetes mellitus with persistent microalbuminuria |
| C109.13 | Type II diabetes mellitus |
| C109.11 | NIDDM - Non-insulin dependent diabetes mellitus |
| 9OLZ.00 | Diabetes monitoring admin.NOS |
| 2G5A.00 | O/E - Right diabetic foot at risk |
| 2BBW.00 | O/E - right eye diabetic maculopathy |
| 2BBX.00 | O/E - left eye diabetic maculopathy |
| 2G5B.00 | O/E - Left diabetic foot at risk |
| 8HBG.00 | Diabetic retinopathy 12 month review |
| 8H7C.00 | Refer, diabetic liaison nurse |
| С109J00 | Insulin treated Type 2 diabetes mellitus |
| 66Af.00 | Patient diabetes education review |
| 66A6.00 | Last hypo. attack |
| ZLA2500 | Seen by diabetic liaison nurse |
| 8Нј0.00 | Referral to diabetes structured education programme |
| 7276.00 | Pan retinal photocoagulation for diabetes |
| C10FL00 | Type 2 diabetes mellitus with persistent proteinuria |
| 8H11.00 | Referral for diabetic retinopathy screening |
| 68AB.00 | Diabetic digital retinopathy screening offered |
| 8Hj4.00 | Referral to DESMOND diabetes structured education programme |
| F420200 | Preproliferative diabetic retinopathy |
| C104.11 | Diabetic nephropathy |
| 8HTk.00 | Referral to diabetic eye clinic |
| 9h400 | Exception reporting: diabetes quality indicators |
| C100.00 | Diabetes mellitus with no mention of complication |
| 2BBL.00 | O/E - diabetic maculopathy present both eyes |
| 66AM.00 | Diabetic - follow-up default |
| 9N2i.00 | Seen by diabetic liaison nurse |

# Protocol for non-interventional studies based on existing data BI Study Number 1245.97

c03856813-11

| Read code | Description |
|-----------|-----------------------------------------------------------|
| C10F.11 | Type II diabetes mellitus |
| M271200 | Mixed diabetic ulcer - foot |
| 2BBR.00 | O/E - right eye preproliferative diabetic retinopathy |
| 66Ae.00 | HbA1c target |
| 2BBS.00 | O/E - left eye preproliferative diabetic retinopathy |
| 8H7f.00 | Referral to diabetes nurse |
| 42c00 | HbA1 - diabetic control |
| M271000 | Ischaemic ulcer diabetic foot |
| 679R.00 | Patient offered diabetes structured education programme |
| F171100 | Autonomic neuropathy due to diabetes |
| 66Am.00 | Insulin dose changed |
| ZL62500 | Referral to diabetes nurse |
| C109700 | Non-insulin dependent diabetes mellitus - poor control |
| F464000 | Diabetic cataract |
| F420z00 | Diabetic retinopathy NOS |
| C10FC00 | Type 2 diabetes mellitus with nephropathy |
| C105.00 | Diabetes mellitus with ophthalmic manifestation |
| 8Hj5.00 | Referral to XPERT diabetes structured education programme |
| 2BBT.00 | O/E - right eye proliferative diabetic retinopathy |
| C10F600 | Type 2 diabetes mellitus with retinopathy |
| M271100 | Neuropathic diabetic ulcer - foot |
| 8H14.00 | Referral to community diabetes specialist nurse |
| 2BBV.00 | O/E - left eye proliferative diabetic retinopathy |
| C104.00 | Diabetes mellitus with renal manifestation |
| 9N0m.00 | Seen in diabetic nurse consultant clinic |
| 9OLB.00 | Attended diabetes structured education programme |
| 9NN9.00 | Under care of diabetes specialist nurse |
| 66Aa.00 | Diabetic diet - poor compliance |
| C107.00 | Diabetes mellitus with peripheral circulatory disorder |
| F372.00 | Polyneuropathy in diabetes |
| 66AJz00 | Diabetic - poor control NOS |

| Read code | Description |
|-----------|---------------------------------------------------------|
| 9N2d.00 | Seen by diabetologist |
| 8H2J.00 | Admit diabetic emergency |
| 2BBF.00 | Retinal abnormality - diabetes related |
| 9OL2.00 | Refuses diabetes monitoring |
| 66Ad.00 | Hypoglycaemic attack requiring 3rd party assistance |
| 8A13.00 | Diabetic stabilisation |
| C10F700 | Type 2 diabetes mellitus - poor control |
| 9N0n.00 | Seen in community diabetes specialist clinic |
| 93C4.00 | Patient consent given for addition to diabetic register |
| 66AJ.11 | Unstable diabetes |
| 9M00.00 | Informed consent for diabetes national audit |
| F420300 | Advanced diabetic maculopathy |
| C10F900 | Type 2 diabetes mellitus without complication |
| 66AJ000 | Chronic hyperglycaemia |
| 66AK.00 | Diabetic - cooperative patient |
| 2G5C.00 | Foot abnormality - diabetes related |
| 66Ap.00 | Insulin treatment initiated |
| 9N0o.00 | Seen in community diabetic specialist nurse clinic |
| 9NN8.00 | Under care of diabetologist |
| ZL62600 | Referral to diabetic liaison nurse |
| C100z00 | Diabetes mellitus NOS with no mention of complication |
| N030100 | Diabetic Charcot arthropathy |
| F381311 | Diabetic amyotrophy |
| TJ23A00 | Adverse reaction to metformin hydrochloride |
| M037200 | Cellulitis in diabetic foot |
| C10FN00 | Type 2 diabetes mellitus with ketoacidosis |
| 66AN.00 | Date diabetic treatment start |
| 8HHy.00 | Referral to diabetic register |
| 2G5H.00 | O/E - Right diabetic foot - ulcerated |
| 2G51000 | Foot abnormality - diabetes related |
| 2G5L.00 | O/E - Left diabetic foot - ulcerated |

## Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1245.97


c03856813-11

| Read code | Description |
|-----------|----------------------------------------------------|
| 66Ak.00 | Diabetic monitoring - lower risk albumin excretion |
| 9OLM.00 | Diabetes structured education programme declined |
| 8CR2.00 | Diabetes clinical management plan |

| Read code | Description |
|-----------|--------------------------------------------------------------|
| C10FK00 | Hyperosmolar non-ketotic state in type 2 diabetes mellitus |
| 66A7100 | Frequency of GP or paramedic treated hypoglycaemia |
| ZV65312 | Dietary counselling in diabetes mellitus |
| C103.00 | Diabetes mellitus with ketoacidotic coma |
| ZRB6.00 | Diabetes wellbeing questionnaire |
| 66AJ200 | Loss of hypoglycaemic warning |
| 9OLK.00 | DESMOND diabetes structured education programme completed |
| C104z00 | Diabetes mellitus with nephropathy NOS |
| F372100 | Chronic painful diabetic neuropathy |
| F3y0.00 | Diabetic mononeuropathy |
| C107.11 | Diabetes mellitus with gangrene |
| F372.11 | Diabetic polyneuropathy |
| 66AL.00 | Diabetic-uncooperative patient |
| 9kL00 | Insulin initiation - enhanced services administration |
| 9OLL.00 | XPERT diabetes structured education programme completed |
| C109400 | Non-insulin dependent diabetes mellitus with ulcer |
| C10D.00 | Diabetes mellitus autosomal dominant type 2 |
| M21yC00 | Insulin lipohypertrophy |
| L180500 | Pre-existing diabetes mellitus, insulin-dependent |
| C109900 | Non-insulin-dependent diabetes mellitus without complication |
| 66A7000 | Frequency of hospital treated hypoglycaemia |
| 8H4e.00 | Referral to diabetes special interest general practitioner |
| C106z00 | Diabetes mellitus NOS with neurological manifestation |
| C102.00 | Diabetes mellitus with hyperosmolar coma |
| K01x100 | Nephrotic syndrome in diabetes mellitus |
| 66AJ300 | Recurrent severe hypos |
| C101z00 | Diabetes mellitus NOS with ketoacidosis |
| G73y000 | Diabetic peripheral angiopathy |
| 66Al.00 | Diabetic monitoring - higher risk albumin excretion |
| ZRbH.00 | Perceived control of insulin-dependent diabetes |
| N030000 | Diabetic cheiroarthropathy |

| Read code | Description |
|-----------|--------------------------------------------------------------|
| 8A12.00 | Diabetic crisis monitoring |
| C105z00 | Diabetes mellitus NOS with ophthalmic manifestation |
| 90LN.00 | Diabetes monitor invitation by SMS (short message service) |
| 8HBH.00 | Diabetic retinopathy 6 month review |
| ZL22500 | Under care of diabetic liaison nurse |
| 9OLF.00 | Diabetes structured education programme completed |
| F35z000 | Diabetic mononeuritis NOS |
| 8H3O.00 | Non-urgent diabetic admission |
| C10FQ00 | Type 2 diabetes mellitus with exudative maculopathy |
| C10G.00 | Secondary pancreatic diabetes mellitus |
| C10F000 | Type 2 diabetes mellitus with renal complications |
| C10F911 | Type II diabetes mellitus without complication |
| C106100 | Diabetes mellitus, adult onset, + neurological manifestation |
| C10FB00 | Type 2 diabetes mellitus with polyneuropathy |
| C10F200 | Type 2 diabetes mellitus with neurological complications |
| 7L10000 | Continuous subcutaneous infusion of insulin |
| 66AG.00 | Diabetic drug side effects |
| 8HLE.00 | Diabetology D.V. done |
| C10FH00 | Type 2 diabetes mellitus with neuropathic arthropathy |
| F372200 | Asymptomatic diabetic neuropathy |
| 9OLG.00 | Attended XPERT diabetes structured education programme |
| C109600 | Non-insulin-dependent diabetes mellitus with retinopathy |
| U60231C | Adverse reaction to metformin hydrochloride |
| 8Hg4.00 | Discharged from care of diabetes specialist nurse |
| F420500 | Advanced diabetic retinal disease |
| 9OL9.00 | Diabetes monitoring deleted |
| M21yC11 | Insulin site lipohypertrophy |
| C10FE00 | Type 2 diabetes mellitus with diabetic cataract |
| 2BBk.00 | O/E - right eye stable treated prolif diabetic retinopathy |
| F372000 | Acute painful diabetic neuropathy |
| 66AO.00 | Date diabetic treatment stopp |

| Read code | Description |
|-----------|------------------------------------------------------------|
| TJ23400 | Adverse reaction to gliclazide |
| 8I3k.00 | Insulin therapy declined |
| C105100 | Diabetes mellitus, adult onset, + ophthalmic manifestation |
| Cyu2.00 | Diabetes mellitus |
| 9OLJ.00 | DAFNE diabetes structured education programme completed |
| C107.12 | Diabetes with gangrene |
| C10zz00 | Diabetes mellitus NOS with unspecified complication |
| 44V3.00 | Glucose tol. test diabetic |
| C10F400 | Type 2 diabetes mellitus with ulcer |
| C10FJ11 | Insulin treated Type II diabetes mellitus |
| 42WZ.00 | Hb. A1C - diabetic control NOS |
| ZLD7500 | Discharge by diabetic liaison nurse |
| C107z00 | Diabetes mellitus NOS with peripheral circulatory disorder |
| C10K.00 | Type A insulin resistance |
| C10A100 | Malnutrition-related diabetes mellitus with ketoacidosis |
| ZV6DA00 | Admitted for commencement of insulin |
| C101000 | Diabetes mellitus, juvenile type, with ketoacidosis |
| 2BB1.00 | O/E - left eye stable treated prolif diabetic retinopathy |
| 9OLH.00 | Attended DAFNE diabetes structured education programme |
| C106.13 | Diabetes mellitus with polyneuropathy |
| R054200 | Gangrene of toe in diabetic |
| C10y.00 | Diabetes mellitus with other specified manifestation |
| C10F711 | Type II diabetes mellitus - poor control |
| C10FL11 | Type II diabetes mellitus with persistent proteinuria |
| U602300 | Insul/oral hypoglyc drugs caus adverse eff therapeut use |
| C10z.00 | Diabetes mellitus with unspecified complication |
| C109C00 | Non-insulin dependent diabetes mellitus with nephropathy |
| C10F100 | Type 2 diabetes mellitus with ophthalmic complications |
| 679L000 | Education in self-management of diabetes |
| C10z100 | Diabetes mellitus, adult onset, + unspecified complication |
| C10FR00 | Type 2 diabetes mellitus with gastroparesis |

| Read code | Description |
|-----------|-------------------------------------------------------------|
| 8Hj3.00 | Referral to DAFNE diabetes structured education programme |
| C10FA00 | Type 2 diabetes mellitus with mononeuropathy |
| C10FD00 | Type 2 diabetes mellitus with hypoglycaemic coma |
| 2G5W.00 | O/E - left chronic diabetic foot ulcer |
| F440700 | Diabetic iritis |
| ZC2CA00 | Dietary advice for type II diabetes |
| C10A.00 | Malnutrition-related diabetes mellitus |
| C10N.00 | Secondary diabetes mellitus |
| R054300 | [D]Widespread diabetic foot gangrene |
| C104100 | Diabetes mellitus, adult onset, with renal manifestation |
| C10N100 | Cystic fibrosis related diabetes mellitus |
| F345000 | Diabetic mononeuritis multiplex |
| C109711 | Type II diabetes mellitus - poor control |
| C107200 | Diabetes mellitus, adult with gangrene |
| C10F500 | Type 2 diabetes mellitus with gangrene |
| 2BBo.00 | O/E - sight threatening diabetic retinopathy |
| C101100 | Diabetes mellitus, adult onset, with ketoacidosis |
| C109712 | Type 2 diabetes mellitus - poor control |
| C107100 | Diabetes mellitus, adult, + peripheral circulatory disorder |
| 8HVU.00 | Private referral to diabetologist |
| C109J12 | Insulin treated Type II diabetes mellitus |
| F381300 | Myasthenic syndrome due to diabetic amyotrophy |
| ZV6DB00 | Admitted for conversion to insulin |
| 8HTi.00 | Referral to multidisciplinary diabetic clinic |
| 66Ae000 | HbA1c target level - IFCC standardised |
| TJ23000 | Adverse reaction to insulins |
| F420700 | High risk proliferative diabetic retinopathy |
| C10F611 | Type II diabetes mellitus with retinopathy |
| 2G5V.00 | O/E - right chronic diabetic foot ulcer |
| C109K00 | Hyperosmolar non-ketotic state in type 2 diabetes mellitus |
| C102100 | Diabetes mellitus, adult onset, with hyperosmolar coma |

| Read code | Description |
|-----------|-------------------------------------------------------------|
| C10FF00 | Type 2 diabetes mellitus with peripheral angiopathy |
| F420800 | High-risk non-proliferative diabetic retinopathy |
| C107400 | NIDDM with peripheral circulatory disorder |
| C10F300 | Type 2 diabetes mellitus with multiple complications |
| 8CP2.00 | Transition of diabetes care options discussed |
| N030011 | Diabetic cheiropathy |
| 66At.00 | Diabetic dietary review |
| C10M.00 | Lipoatrophic diabetes mellitus |
| 9M10.00 | Informed dissent for diabetes national audit |
| C10FP00 | Type 2 diabetes mellitus with ketoacidotic coma |
| C109611 | Type II diabetes mellitus with retinopathy |
| C10FG00 | Type 2 diabetes mellitus with arthropathy |
| C109J11 | Insulin treated non-insulin dependent diabetes mellitus |
| C101y00 | Other specified diabetes mellitus with ketoacidosis |
| C109411 | Type II diabetes mellitus with ulcer |
| 8I2S.00 | Glitazones contraindicated |
| C109000 | Non-insulin-dependent diabetes mellitus with renal comps |
| C109100 | Non-insulin-dependent diabetes mellitus with ophthalm comps |
| C106y00 | Other specified diabetes mellitus with neurological comps |
| TJ23.00 | Adverse reaction to insulins and antidiabetic agents |
| 9h43.00 | Excepted from diabetes qual indicators: service unavailable |
| C106.11 | Diabetic amyotrophy |
| TJ23z00 | Adverse reaction to insulins and antidiabetic agents NOS |
| C104y00 | Other specified diabetes mellitus with renal complications |
| C109612 | Type 2 diabetes mellitus with retinopathy |
| C109212 | Type 2 diabetes mellitus with neurological complications |
| C109200 | Non-insulin-dependent diabetes mellitus with neuro comps |
| C106000 | Diabetes mellitus, juvenile, + neurological manifestation |
| ZRB4.00 | Diabetes clinic satisfaction questionnaire |
| C109412 | Type 2 diabetes mellitus with ulcer |
| ZRB5.11 | DTSQ - Diabetes treatment satisfaction questionnaire |

| Read code | Description |
|-----------|--------------------------------------------------------------|
| C109E00 | Non-insulin depend diabetes mellitus with diabetic cataract |
| 8I2P.00 | Sulphonylureas contraindicated |
| C109B00 | Non-insulin dependent diabetes mellitus with polyneuropathy |
| C109E11 | Type II diabetes mellitus with diabetic cataract |
| 8HKE.00 | Diabetology D.V. requested |
| C10yz00 | Diabetes mellitus NOS with other specified manifestation |
| C109C12 | Type 2 diabetes mellitus with nephropathy |
| C109500 | Non-insulin dependent diabetes mellitus with gangrene |
| С109Н00 | Non-insulin dependent d m with neuropathic arthropathy |
| C109D00 | Non-insulin dependent diabetes mellitus with hypoglyca coma |
| C109011 | Type II diabetes mellitus with renal complications |
| C109300 | Non-insulin-dependent diabetes mellitus with multiple comps |
| U602312 | Adverse reaction to insulins |
| C10zy00 | Other specified diabetes mellitus with unspecified comps |
| U602311 | Adverse reaction to insulins and antidiabetic agents |
| TJ23500 | Adverse reaction to glipizide |
| 66Ar.00 | Insulin treatment stopped |
| C109H11 | Type II diabetes mellitus with neuropathic arthropathy |
| 889A.00 | Diab mellit insulin-glucose infus acute myocardial infarct |
| C109H12 | Type 2 diabetes mellitus with neuropathic arthropathy |
| 9NiC.00 | Did not attend DAFNE diabetes structured education programme |
| 66AQ100 | Declined consent for diabetes year of care programme |
| C10yy00 | Other specified diabetes mellitus with other spec comps |
| C10F311 | Type II diabetes mellitus with multiple complications |
| C109E12 | Type 2 diabetes mellitus with diabetic cataract |
| C108y00 | Other specified diabetes mellitus with multiple comps |
| TJ23300 | Adverse reaction to glibenclamide |
| C109511 | Type II diabetes mellitus with gangrene |
| C10y100 | Diabetes mellitus, adult, + other specified manifestation |
| C10N000 | Secondary diabetes mellitus without complication |
| 66As.00 | Diabetic on subcutaneous treatment |

| Read code | Description |
|-----------|--------------------------------------------------------------|
| 66At100 | Type II diabetic dietary review |
| C109012 | Type 2 diabetes mellitus with renal complications |
| C109D12 | Type 2 diabetes mellitus with hypoglycaemic coma |
| U602316 | Adverse reaction to gliclazide |
| C102z00 | Diabetes mellitus NOS with hyperosmolar coma |
| C109512 | Type 2 diabetes mellitus with gangrene |
| C109F00 | Non-insulin-dependent d m with peripheral angiopath |
| C109C11 | Type II diabetes mellitus with nephropathy |
| C103z00 | Diabetes mellitus NOS with ketoacidotic coma |
| 9N1o.00 | Seen in multidisciplinary diabetic clinic |
| C109G00 | Non-insulin dependent diabetes mellitus with arthropathy |
| C105y00 | Other specified diabetes mellitus with ophthalmic complicatn |
| C109F11 | Type II diabetes mellitus with peripheral angiopathy |
| C10FM11 | Type II diabetes mellitus with persistent microalbuminuria |
| C10F411 | Type II diabetes mellitus with ulcer |
| 66Au.00 | Diabetic erectile dysfunction review |
| 66Av.00 | Diabetic assessment of erectile dysfunction |
| Cyu2000 | Other specified diabetes mellitus |
| C109B11 | Type II diabetes mellitus with polyneuropathy |
| C10F011 | Type II diabetes mellitus with renal complications |
| C103y00 | Other specified diabetes mellitus with coma |
| C109211 | Type II diabetes mellitus with neurological complications |
| ZRB4.11 | CSQ - Diabetes clinic satisfaction questionnaire |
| 3883.00 | Diabetes treatment satisfaction questionnaire |
| 8IAs.00 | Diabetic dietary review declined |
| 2BBr.00 | Impaired vision due to diabetic retinopathy |
| TJ23900 | Adverse reaction to tolbutamide |
| C10FB11 | Type II diabetes mellitus with polyneuropathy |
| C109D11 | Type II diabetes mellitus with hypoglycaemic coma |
| C109111 | Type II diabetes mellitus with ophthalmic complications |
| C109F12 | Type 2 diabetes mellitus with peripheral angiopathy |

## c03856813-11

| Read code | Description |
|-----------|-------------------------------------------------------------|
| C10A000 | Malnutrition-related diabetes mellitus with coma |
| C103100 | Diabetes mellitus, adult onset, with ketoacidotic coma |
| C109A00 | Non-insulin dependent diabetes mellitus with mononeuropathy |
| 8HME.00 | Listed for Diabetology admissn |
| C10FA11 | Type II diabetes mellitus with mononeuropathy |
| U60231B | Adverse reaction to tolbutamide |
| U60231E | Adverse reaction to insulins and antidiabetic agents NOS |
| Cyu2300 | Unspecified diabetes mellitus with renal complications |
| 8HgC.00 | Discharged from diabetes shared care programme |
| 66AQ000 | Unsuitable for diabetes year of care programme |
| C10F111 | Type II diabetes mellitus with ophthalmic complications |
| TJ23B00 | Adverse reaction to glucagon |
| C109G11 | Type II diabetes mellitus with arthropathy |
| U602315 | Adverse reaction to glibenclamide |
| C109G12 | Type 2 diabetes mellitus with arthropathy |
| C109A11 | Type II diabetes mellitus with mononeuropathy |
| C10K000 | Type A insulin resistance without complication |
| U60231A | Adverse reaction to tolazamide |
| C108z00 | Unspecified diabetes mellitus with multiple complications |
| C109112 | Type 2 diabetes mellitus with ophthalmic complications |
| U602318 | Adverse reaction to gliquidone |
| TJ23200 | Adverse reaction to chlorpropamide |
| C10FE11 | Type II diabetes mellitus with diabetic cataract |
| U602317 | Adverse reaction to glipzide |
| C10G000 | Secondary pancreatic diabetes mellitus without complication |
| ZRB6.11 | DWBQ - Diabetes wellbeing questionnaire |
| C10F211 | Type II diabetes mellitus with neurological complications |
| C10E512 | Insulin-dependent diabetes mellitus with ulcer |
| C10FD11 | Type II diabetes mellitus with hypoglycaemic coma |
| SL23100 | Biguanide poisoning |
| Kyu0300 | Glomerular disorders in diabetes mellitus |

## Boehringer Ingelheim Protocol for non-interven


## Protocol for non-interventional studies based on existing data BI Study Number 1245.97

c03856813-11

| Read code | Description |
|-----------|--------------------------------------------------------------|
| C10A500 | Malnutritn-relat diabetes melitus wth periph circul completn |
| C10FC11 | Type II diabetes mellitus with nephropathy |
| 66Aw.00 | Insulin dose |
| TJ23800 | Adverse reaction to tolazamide |

## ANNEX 4. CODES TO IDENTIFY EXPOSURE VARIABLES

| No. | Variable | ATC codes <sup>3</sup> | Time-dependent<br>(T) / fixed at<br>cohort entry (F) | How the effect of variable is accounted for <sup>1</sup> |
|---|---|---|---|---|
| 1 | AT / ITT: Empagliflozin | Empagliflozin A10BK03 (current), A10BX12 (previous) | T/F | Е |
| 2 | AT / ITT: DPP-4 inhibitor | DPP-4 inhibitors ATC beginning with A10BH Fixed-dose combinations Will be identified from ATC class A10BD | T/F | E |
| 3 | AT / ITT, FDCM <sup>2</sup> : empagliflozin | | T/F | Е |
| 4 | AT / ITT, FDCM <sup>2</sup> : DPP-4 inhibitor | | T / F | Е |
| 5 | Empagliflozin current use | | Т | Е |
| 6 | Empagliflozin: cumulative duration of exposure | | Т | Е |
| 7 | Empagliflozin: cumulative dosage of exposure | | Т | Е |
| 8 | Empagliflozin: time since last dose | | Т | Е |
| | Other OAD treatments | | | |
| 9 | Metformin | ATC beginning with A10BA | Т | PS / A / VS, RS,<br>TV, SG |
| 10 | Sulphonylureas | ATC beginning with A10BB | Т | PS / A / VS, RS,<br>TV |

| No. | Variable | ATC codes <sup>3</sup> | Time-dependent<br>(T) / fixed at<br>cohort entry (F) | How the effect of variable is accounted for <sup>1</sup> |
|---|---|---|---|---|
| 11 | Insulin | ATC beginning with A10A | Т | PS / A / VS, RS,<br>TV |
| 12 | Thiazolidinediones | ATC beginning with A10BG | Т | PS / A / VS, RS,<br>TV |
| 13 | Alpha glucosidase inhibitors | ATC beginning with A10BF | Т | PS / A / VS, RS,<br>TV |
| 14 | GLP-1 agonists | Will be identified<br>from ATC classes<br>A10BJ and A10BX | Т | PS / A / VS, RS,<br>TV |
| 15 | Other blood glucose lowering drugs, excluding insulins | ATC beginning with A10BX that is not included elsewhere | | |
| 16 | Treatment complexity<br>(mono, dual and triple<br>combination therapy) | | Т | PS / A / VS, RS,<br>TV |
| 17 | Switch or add-on | | Т | PS / A / VS, RS,<br>TV |
| | Exclusion / Censoring | | | |
| 18 | DPP-4 (Linagliptin) and<br>Empagliflozin | A10BD19 | Т | Censoring /<br>Exclusion |
| 19 | Discontinuation of primary exposure | | Т | Censoring |
| 20 | Switch to other SGLT-2 inhibitor use | A10BK02,<br>A10BX11,<br>A10BK01,<br>A10BX09,<br>A10BK04,<br>A10BD16,<br>A10BD15,<br>A10BD23 | Т | Censoring /<br>Exclusion |

## **Boehringer Ingelheim**

## 

## Protocol for non-interventional studies based on existing data BI Study Number 1245.97

c03856813-11

| No. | Variable | ATC codes <sup>3</sup> | Time-dependent<br>(T) / fixed at<br>cohort entry (F) | How the effect of variable is accounted for <sup>1</sup> |
|---|---|---|---|---|
| 21 | Use of fixed-dose<br>combinations of SGLT-2<br>inhibitors with DPP-4<br>inhibitors | Identified from<br>ATC class A10BD | Т | Censoring /<br>Exclusion |

<sup>&</sup>lt;sup>1</sup> E – Exposure, A – adjusted in the Cox model, VS – potential confounder and will be adjusted for using variable selection, PS – one of the PS matching variable at baseline, TV – time-varying confounder and adjusted for in MSM, RS – defines the risk set in NCC, SG – used as a subgroup in stratified analyses, /- and/or

<sup>2</sup> FDCM – Fixed-dose combination with metformin

<sup>3</sup> New drugs will be included in the variable definitions if they become available during the study period.

## ANNEX 5. CODES TO IDENTIFY THE OUTCOME VARIABLES

The codes will be updated for the data applications.

| No. | Variable | ICD-10 / ICD-<br>O-3 codes | READ codes | Outcome /<br>Censoring<br>variable | Analyses <sup>1</sup> |
|---|---|---|---|---|---|
| 1 | Urinary Tract cancer (malignant and carcinoma in situ) | C64-C68<br>D09.0, D09.1 | Byu9, B837,<br>B83z, B4A,<br>B49 | Outcome | D, P, S, F,<br>NCC, MSM<br>Sens |
| 2 | Bladder cancer (malignant and carcinoma in situ) | C67, D09.0 | B49, B837,<br>selected<br>BB4 codes | Outcome | D, P, S, F, Sens |
| 3 | Renal cancer (malignant) | C64, C65 | B4A0, B4A1 | Outcome | D, P, S, F, Sens |
| 4 | Other urinary tract<br>cancer (non-renal,<br>non-bladder cancers) –<br>sensitivity (malignant) | C66,C68 | Byu9 | Sensitivity outcome | D, Sens |
| 5 | Urinary Tract cancers<br>from GP data (CPRD<br>only) – sensitivity | | Byu9, B837,<br>B83z, B4A,<br>B49 | Sensitivity outcome | Sens |
| 6 | Urinary tract<br>neoplasms of uncertain<br>or unknown behaviour<br>- sensitivity | D41 | B917, B91z,<br>BA04 | Sensitivity outcome | Sens |
| | Censoring variables | | | | |
| 7 | Other non-UT cancers | C00-C99, D00-<br>09 (excl. C64-<br>68, D09.0,<br>D09.1) | B (excl.<br>Byu9, B837,<br>B83z, B4A,<br>B49, B49,<br>B837,<br>selected<br>BB4 codes) | Censoring | |
| 8 | End of study period | | | Censoring | |
| 9 | End of GP practice coverage | | | Censoring | |
| 10 | Use of other SGLT-2 (since start of follow-up) | | | Censoring | |
| 11 | Use of fixed-dose combinations of | | | Censoring | |

## Boehringer Ingelheim


Protocol for non-interventional studies based on existing data BI Study Number 1245.97

c03856813-11

| No. | Variable | ICD-10 / ICD-<br>O-3 codes | READ codes | Outcome /<br>Censoring<br>variable | Analyses <sup>1</sup> |
|---|---|---|---|---|---|
| | SGLT-2 inhibitors with DPP-4 inhibitors | | | | |
| 12 | Patient transfer | | | Censoring | |
| 13 | End stage renal disease / renal dialysis | | | Censoring | |
| 14 | All-cause mortality (excluding UT cancer mortality) | | | Censoring | |
| 15 | Discontinuation of primary exposure | | | Censoring for as-treated analysis | |
| 16 | UT cancer characteristics (based on staging, TNM codes, etc) | | | Sensitivity<br>outcome /<br>descriptive | D, Sens |

 $<sup>1\</sup> D = Descriptive,\ P = Primary\ ,\ S = secondary,\ F = further,\ Sens = sensitivity,\ NCC = Nested-case-control,\ MSM-marginal\ structural\ models$ 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## ANNEX 6. COVARIATES TO BE CONSIDERED FOR INCLUSION IN THE PROPENSITY SCORE MODEL.

| No. | Variable |
|-----|----------------------------------------------|
| | Socio-demographic variables |
| 1 | Age |
| 2 | Sex |
| 3 | Socioeconomic status |
| 4 | Calendar year of index date |
| 5 | Duration of look-back period |
| 6 | Duration of treated diabetes at index date |
| | Diabetic complications |
| 7 | Diabetic retinopathy or diabetic maculopathy |
| 8 | Diabetic nephropathy |
| 9 | Diabetic neuropathy |
| 10 | Peripheral vascular disease |
| 11 | Diabetic lower limb severe complications |
| | Urinary tract related comorbidities |
| 12 | Kidney or genitourinary stones |
| 13 | Prior history of UTI or pyelonephritis |
| 14 | Liver disease |
| 15 | eGFR |
| 16 | Renal impairment |
| 17 | Prior ICU admission |
| 18 | Pancreatitis |

## Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1245.97


c03856813-11

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 19 | BMI (when available) |
|----|------------------------------------------------|
| 20 | Smoking (when available) |
| 21 | Alcohol use (when available) |
| 22 | HbA1c (when available) |
| 23 | Albuminuria testing |
| | Cardiovascular Diseases |
| 24 | Congestive heart failure |
| 25 | Blood pressure measurements |
| 26 | Hypertension |
| 27 | Stroke |
| 28 | Myocardial infarction |
| 29 | Autoimmune disease |
| 30 | COPD |
| 31 | Time since first diabetes diagnosis |
| | Other non-diabetes medications |
| 32 | Antihypertensives/diuretics |
| 33 | Non-steroidal anti-inflammatory drugs (NSAIDs) |
| 34 | Oral steroids |
| 35 | Statins, fibrates |
| 36 | Lipid modifying agents |
| 37 | Zoledronic acid |
| 38 | Antibiotics |
| 39 | Other drugs |
| _ | |

BMI=body mass index; COPD=chronic obstructive pulmonary disease; eGFR=estimated glomerular filtration rate; HbA1c=glycated haemoglobin A1c; HF=heart failure; ICU=intensive care unit; MSM=marginal structural model; NCC=nested case-control; PS=propensity score; UTI=urinary tract infection.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **SIGNATURE**

#### PRINCIPAL INVESTIGATOR SIGNATURE

Study Title: Post-authorisation safety study to assess the risk of urinary tract

malignancies in relation to Empagliflozin exposure in patients with type 2

diabetes: a multi-database European study

Trial Number: 1245.97

Affiliation:

Study protocol version: 8.0

I herewith certify that I agree to content of Study protocol version 8.0 and to all documents referenced in the study protocol version 8.0.

Company)

| Date: 02-Jun | -2023 | | |
|---|---|---|---|
| Name: | | Signature: | Signer Name Signing Reason: Lapprove this document Signing Time: 02-Jun-2023 12:05:57 AM PDI |



#### APPROVAL / SIGNATURE PAGE

Document Number: c03856813 Technical Version Number:11.0

Document Name: 1245-0097-clinical-trial-protocol

**Title:** Post-authorisation safety study to assess the risk of urinary tract malignancies in relation to empagliflozin exposure in patients with type 2 diabetes: a multi-database European study

## Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Approval-EU Qualified Person<br>Pharmacovigilance | | 15 Jun 2023 14:04 CEST |
| Verification-Paper Signature<br>Completion | | 15 Jun 2023 14:13 CEST |
| Approval | | 15 Jun 2023 15:02 CEST |
| Approval-On behalf of or VP | | 15 Jun 2023 15:21 CEST |
| Approval | | 15 Jun 2023 16:57 CEST |
| Approval-Team Member Drug<br>Safety | | 19 Jun 2023 17:28 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c03856813Technical Version Number: 11.0

## (Continued) Signatures (obtained electronically)

| Meaning of Signature Signed by Date Signed |
|--------------------------------------------|
|--------------------------------------------|